

A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of RA101495 in Subjects with Generalized Myasthenia Gravis

Statistical Analysis Plan Version: Date of Statistical Analysis Plan:

Version 1.0 Version 2.0 05Nov2018 05Mar2020

### SIGNATURE PAGE

| | :Orsor V |
|---|---|
| Date | Prepared by:, PhD Senior Statistical Consultant |
| | Prepared by:, PhD Senior Statistical Consultant Prepared by:, PhD Senior Statistical Consultant |
| Date | Reviewed and Approved by: |
| Date Date Date Leannot be used to support any many many many many many many many | Senior Director, Clinical Research Ra Pharmaceuticals, Inc. |
| Date Support | Reviewed and Approved by: MD FACC Chief Medical Officer, Ra Pharmaceuticals, Inc. |
| Leannot be us | |


#### **DOCUMENT HISTORY**

| | Version | Author | Description |
|---|---|---|---|
| | 1.0 | | Original Version |
| | 2.0 | | Updated to include Extension Period analyses |
| This document | i cannot be use | ato support any mark | Original Version Updated to include Extension Period analyses in appendix Description Updated to include Extension Period analyses in appendix Description Updated to include Extension Period analyses in appendix Description Updated to include Extension Period analyses in appendix Description Description Updated to include Extension Period analyses in appendix Description Description Updated to include Extension Period analyses in appendix Description Desc |
| | CONF | IDENTIAL | |

### Table of Contents

| 1 | INTR | RODUCTION | 10 |
|---|-------|----------------------------------------------------|-------------|
| 2 | STUI | DY SUMMARY | 10 |
| | 2.1 | STUDY OBJECTIVES | 10 |
| | 2.2 | STUDY DESIGN | 13 |
| | 2.2.1 | Number of Subjects | :0.12 |
| | 2.2.2 | Randomization and Blinding Procedures | 12 |
| | 2.3 | Number of Subjects | 12 |
| | 2.3.1 | Physical Examination | 13 |
| | 2.3.2 | Vital Signs | 13 |
| | 2.3.3 | Electrocardiogram | 13 |
| | 2.3.4 | Laboratory Assessments | 13 |
| | 2.3.6 | Immunogenicity | 15 |
| | 2.4 | Efficacy Assessments | 16 |
| | 2.4.1 | Quantitative Myasthenia Gravis Score | 16 |
| | 2.4.2 | Myasthenia Gravis Activities of Daily Living Score | 16 |
| | 2.4.3 | Myasthenia Gravis Quality of Life | 17 |
| | 2.4.4 | MG Composite | 17 |
| | 2.5 | | |
| | 2.5 | Pharmacodynamic Assessments | |
| C | 2.7 | Rescue Therapy | |
| | 2.8 | Schedule of Assessments | |
| 3 | | ΓISTICAL METHODS | |
| J | 3.1 | General Methods | |
| | | | age 4 of 61 |

CONFIDENTIAL


| 3.1.1 | Computing Environment | 31 |
|---|---|---|
| 3.1.2 | Reporting of Numerical Values | 31 |
| 3.1.3 | Baseline Value and Change from Baseline | 31 |
| 3.2 | Handling of Missing Values | 32 |
| 3.2.1 | Efficacy Endpoints: Main Portion | 32 |
| 3.2.2 | Efficacy Endpoints: Extension Portion | |
| 3.2.3 | Safety, PK and PD Endpoints | |
| 3.3 | Efficacy Endpoints: Main Portion Efficacy Endpoints: Extension Portion Safety, PK and PD Endpoints Analysis Populations Intention-to-Treat Population Modified ITT Population Per Protocol Population Safety Population RA101495 Safety Population | 34 |
| 3.3.1 | Intention-to-Treat Population | 34 |
| 3.3.2 | Modified ITT Population | 34 |
| 3.3.3 | Per Protocol Population | 34 |
| 3.3.4 | Safety Population | 34 |
| 3.3.5 | RA101495 Safety Population | 35 |
| 3.3.6 | Pharmacokinetic Population | 35 |
| 3.3.7 | Pharmacodynamic Population | 35 |
| 3.4 | Combining RA101495 Data Across Study Portions | 35 |
| 3.5 | Efficacy Endpoints | 36 |
| 3.5.1 | À. • | 36 |
| 3.5.2 | Secondary Efficacy Endpoints | 36 |
| 3.6 | Pharmacodynamic Endpoints | 36 |
| IMERIT 3.7 | Exploratory Endpoints | 36 |
| 3.5.2<br>3.5.2<br>3.5.2<br>3.7<br>3.8<br>7his document 3.8<br>3.8.1 | Patient Disposition and Evaluability | 37 |
| 3.8.1 | Patient Disposition | 37 |
| 3.8.2 | Protocol Deviations | 37 |

| 3.9 | Demographics and Baseline Characteristics |
|--------|-----------------------------------------------------------|
| 3.9.1 | Demographics |
| 3.9.2 | Medical History |
| 3.9.3 | Demographics |
| 3.10 | Prior and Concomitant Medications |
| 3.11 | MG Specific Prior and Concomitant Medications |
| 3.12 | Exposure to Study Treatment |
| 3.13 | Prior and Concomitant Medications |
| 3.13. | 1 Adverse Events |
| 3.13.2 | 2 Clinical Laboratory Evaluation |
| 3.13.3 | 3 Vital Signs and Other Physical Findings |
| 3.13.4 | 4 ECG |
| 3.13.5 | 5 Physical Examination |
| 3.14 | Efficacy Analyses |
| 3.14. | Primary Efficacy Endpoint Analysis |
| 3.14.2 | 2 Secondary Efficacy Endpoints Analysis |
| 3.15 | Controlling for Multiplicity |
| 3.15. | Additional Analyses of Primary and Secondary Endpoints 50 |
| 3.15 | Pharmacodynamic Endpoints Analysis |
| 3.15.3 | 3 Pharmacokinetic Endpoints Analysis 54 |
| 3.15.4 | 4 Exploratory Endpoints Analysis |
| 3.16 | Additional Analyses55 |
| 3.16. | 1 Rescue Therapy55 |
| 3.17 | Interim Analysis |
| CC | ONFIDENTIAL |

| 3.18 | Timing of Primary Analysis | 56 |
|---|---|---|
| 3.19 | Sample Size Considerations | 56 |
| 3.20 | Replacement of Subjects | 56 |
| 3.21 | Protocol Violations | 56 <sub>ili</sub> dil <sup>oli</sup> |
| 4 Refer | rences | 56 |
| 5 Appe | Sample Size Considerations | 2.58 |
| 6 Appe | ndix 2: Analyses Including Data After Day E84 | 59 |
| 6.1 | Additional Analysis Population: Extension Population Disposition | 59 |
| 6.2 | Disposition | 59 |
| 6.3 | Subject Switching From 0.1 mg/kg to 0.3 mg/kg | 59 |
| 6.4 | Exposure | 59 |
| 6.5 | Exposure Efficacy Endpoints Safety Endpoints Adverse Events | 60 |
| 6.6 | Safety Endpoints | 61 |
| 6.6.1 | Adverse Events | 61 |
| 6.6.2 | ~************************************* | 61 |
| This document cannot be | Jused to Support all. | |
| This docu | | |


### LIST OF ABBREVIATIONS

| LIST OF ABBREVIATION | | |
|---|---|---|
| Abbreviation | Full Term | , variations thereof. |
| ADA | anti-drug antibody | ei/eo |
| AE | adverse event | Eille |
| ALP | alkaline phosphatase | ijon <sup>3</sup> |
| ALT | alanine aminotransferase | ajiali |
| ANCOVA | analysis of covariance | 10. |
| aPTT/APTT | activated partial thromboplastin time | )* |
| AST | aspartate aminotransferase | |
| BMI | body mass index | |
| BUN | blood urea nitrogen | |
| C5 | complement component 5 | |
| cm | centimeter | |
| C <sub>max</sub> | maximum plasma concentration | |
| CPK | creatine phosphokinase | |
| CRP | C-reactive protein | |
| CSR | clinical study report | |
| CTCAE | Common Terminology Criteria for Adverse Events | |
| ECG | electrocardiogram | |
| eCRF | electronic case report form | |
| GGT | gamma-glutamyl transferase | |
| HR | heartrate | |
| ICF | informed consent form | |
| ICH | International Conference on Harmonization | |
| INR X | international normalized ratio | |
| ISR | injection site reaction | |
| ITT 5 <sup>N</sup> | intent-to-treat | |
| kg | kilogram | |
| LOCF 5 | last observation carried forward | |
| MCV | mean corpuscular volume | |
| MedDRA | Medical Dictionary for Regulatory Activities | |
| MG-ADL | myasthenia gravis activities of daily living | |
| mg | milligram | |
| mITT | modified intent-to-treat | |
| MMRM | mixed model repeated measures | |
| NCI | National Cancer Institute | |
| PD | pharmacodynamics | |
| PK | pharmacokinetics | |


| DATE | 1 , 11 11 . | |
|---|---|---|
| PNH | paroxysmal nocturnal hemoglobinuria | |
| PT | prothrombin time | atiations thereof. |
| PT | preferred term | - exec |
| PTT | partial thromboplastin time | Sille |
| QMG | quantitative myasthenia gravis | *ion3 |
| QOL | quality of life | ailat |
| SAE | serious adverse event | 70 |
| SAP | statistical analysis plan | |
| SC | statistical analysis plan subcutaneously system organ class sheep red blood cell | |
| SOC | system organ class | |
| sRBC | sheep red blood cell | |
| TEAE | treatment-emergent adverse event | |
| $t_{max}$ | time to corresponding Cmax | |
| ULN | upper limit of normal | |
| WBC | white blood cell | |
| TEAE tmax ULN WBC | Refind authoric Amarke in a string in the st | |
| CONFIDENTIAL | | |

#### 1 INTRODUCTION

ions of variations thereof. Ra Pharmaceuticals, Inc. is developing RA101495, a subcutaneously (SC) selfadministered 15-amino acid cyclic peptide that binds to, and inhibits the cleavage of, complement component 5 (C5).

Study RA101495-02.201 is a multicenter, randomized, double-blind, placebocontrolled study to evaluate the safety, tolerability, and preliminary efficacy of RA101495 in subjects with gMG. The planned enrollment is approximately 36 subjects.

Subjects will be randomized in a 1:1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495, 0.3 mg/kg RA101495, or matching placebo.

This Statistical Analysis Plan (SAP) describes data-handling and statistical procedures to be used for the analysis and reporting of efficacy and safety data collected under Study RA101495-02.201 (version 2.0 19 October 2017) and presented in the clinical study report (CSR). The methods are based on those presented in Section 12 of the study protocol. Any post-hoc or exploratory analyses not specified in this SAP will be identified as such when they are presented in the CSR. This SAP has been developed and finalized prior to locking the clinical database for the Main Portion of the study.

The analyses involving the Main Portion and the first 12 Weeks of the Extension Portion (i.e., through study day E84) will be included in the main section of this SAP document. Analyses involving the whole study, including the entire open-label Extension Portion beyond study day E84 will be in the appendix of this document. The reason for the analyses being separated into two distinct sections of the SAP document is to allow for the analysis methods relating to the randomized double-blind portion of the study to be finalized while allowing for future modifications to the analyses of the open-label Extension Portion (note: this method is consistent with the study protocol in that the schedule of assessments after day E84 is in the Protocol Appendix).

This SAP was written in accordance with the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled "Guidance for Industry: Statistical Principles for Clinical Trials" and the most recent ICH-E3 Guideline, entitled "Guidance for Industry: Structure and Content of Clinical Study Reports."

#### STUDY SUMMARY

#### 2.1 STUDY OBJECTIVES

The objectives of the study are:

• To assess the safety and tolerability of RA101495 in subjects with gMG  To assess preliminary efficacy of RA101495 in subjects with gMG

Subjects will be randomized in a 1:1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495, 0.3 mg/kg RA101495, or matching placebo. Randomization will be stratified based on the screening QMG Score (≤ 17 versus ≥ 18).

The Main Portion of the study includes a Screening of the clinic weels.

followed by visits at Week 4 (Day 29), Week 8 (Day 57), and Week 12 (Day 84) to evaluate safety, tolerability, and preliminary efficacy. Additional assessments will include quality of life (QOL) questionnaires, biomarker samples, pharmacokinetics, pharmacodynamics, and optional pharmacogenomics. Safety assessments will include physical examinations, vital signs, ECGs, clinical laboratory tests, adverse events (AEs), and immunogenicity.

Randomized subjects will receive 0.1 mg/kg RA101495, 0.3 mg/kg RA101495, or matching placebo administered SC at the Day 1 visit. Following in-clinic education and training, all subjects will self-inject daily SC doses of blinded study drug, according to randomized treatment allocation, for the subsequent 12 weeks. A singleuse, disposable, injection device will be provided for use during the study.

At the conclusion of the Treatment Period in the Main Portion of the study, all subjects will have the option to receive RA101495 in the Extension Portion of the study provided they meet the Extension Portion selection criteria (Protocol Section 8.3). Subjects assigned to a RA101495 treatment arm during the Main Portion of the study will continue to receive the same dose of study drug during the Extension Portion. Subjects assigned to the placebo arm during the Main Portion of the study will be randomized in a 1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495 or 0.3 mg/kg RA101495. Assessments and visits during the first 12 weeks of the Extension Portion will be identical to the Main Portion of the study for all subjects to ensure appropriate monitoring of subjects transitioning from placebo to active treatment and to maintain blinding of treatment assignment. The study will remain double-blinded during the Extension Portion until after the data from the Main Portion of the study have been cleaned, locked, and unblinded.

Figure 1 provides an illustration of the study design.




Figure 1: Design of RA101495-02.201

#### 2.2.1 Number of Subjects

Approximately 36 subjects will be randomized (i.e., 12 per treatment arm):

### 2.2.2 Randomization and Blinding Procedures

Subjects who meet all entry criteria will be randomized in a 1:1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495, 0.3 mg/kg RA101495, or matching placebo. Subjects will be assigned to study arms in a blinded fashion using a computerized randomization algorithm. Randomization will be stratified based on the screening QMG Score ( $\leq$  17 versus  $\geq$  18).

Subjects assigned to a RA101495 treatment arm during the Main Portion of the study will continue to receive the same dose of study drug during the Extension Portion. Subjects assigned to the placebo arm during the Main Portion of the study will be randomized in a 1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495 or 0.3 mg/kg RA101495. This randomization will occur at the screening visit when the subject is initially randomized to the Main Portion of the study.

This is a double-blind study. Subjects and study staff will remain blinded to treatment assignments until after the data from the Main Portion of the study have been cleaned, locked, and unblinded.

The procedure for emergency unblinding of study drug treatment for an individual subject is discussed in protocol section 11.3.3.

### 2.3 Safety Assessments

Safety assessments will include physical examinations, vital signs, ECGs, clinical laboratory tests, AEs, and immunogenicity.


#### 2.3.1 **Physical Examination**

any extensions or variations thereof. A full physical examination will be performed on all subjects at the Screening visit and will include the following assessments:

- General inspection
- Examination of the injection site and draining nodes
- Head/ears/eyes/nose/throat examination
- Mucosal examination
- Cardiac examination
- Auscultation of lungs
- Abdominal examination (liver, spleen, and lower abdomen)
- Musculoskeletal assessment
- Neurological assessment

Any abnormalities found will be recorded in the electronic case report form (eCRF).

At all other study visits, the physical examination will be symptom-directed.

#### 2.3.2 Vital Signs

Vital signs (Heart Rate (HR), body temperature, and blood pressure) will be measured in the sitting position. Blood pressure may be measured manually or by automated device, preferably using the non-dominant arm. The same measurement technique should be used throughout the study for all the subjects.

#### 2.3.3 Electrocardiogram

12-lead ECGs will be assessed as normal or abnormal by the investigator; any abnormal findings will be described in the eCRF and the investigator will assess clinical significance. The ECG recording strip will be signed and dated by the investigator and stored in the medical records.

ECGs should be performed prior to blood draws when both assessments are required at the same visit.

### 2.3.4 Laboratory Assessments

y, nematology, coagulation (for the control laboratory are to be performed by a central laboratory set the study database. Values from local laboratories may be used to determine eligibility for study enrollment and as the basis for clinical decisions Safety laboratory tests for this study [chemistry, hematology, coagulation (for applicable subjects), and urinalysis] are to be performed by a central laboratory, and only values from the central laboratory are to be entered into the laboratory section of

> 

### 2.3.4.1 Hematology, Chemistry, and Coagulation

A variations thereof. Hematology, chemistry, and coagulation analytes that will be assessed during the study are identified in Table 1. Coagulation tests should only be performed in subjects receiving anticoagulant therapy.

Table 1: Clinical Chemistry, Hematology, and Coagulation Analytes

| Clinical Chemistry | Hematology |
|---|---|
| Alanine aminotransferase (ALT) | Hematocrit Hemoglobin Mean corpuscular volume (MCV) |
| Albumin | Hemoglobin |
| Alkaline phosphatase (ALP) | Mean corpuscular volume (MCV) |
| Amylase | Platelet count |
| Aspartate aminotransferase (AST) | White blood cell (WBC) count and differential (%) |
| Bicarbonate | <ul> <li>basophils</li> <li>eosinophils</li> <li>lymphocytes</li> <li>monocytes</li> <li>neutrophils</li> </ul> |
| Bile acids | • eosinophils |
| Bilirubin (total, direct, and indirect) | • lymphocytes |
| Blood urea nitrogen (BUN) | • monocytes |
| Calcium | • neutrophils |
| Chloride | Coagulation |
| Creatinine | International normalized ratio (INR)/prothrombin |
| Gamma-glutamyl transferase (GGT) | time (PT) |
| Glucose | Fibrinogen |
| Lipase | Partial thromboplastin time (PTT) or activated |
| Potassium | partial thromboplastin time (aPTT) |
| Sodium | Other |
| Total protein | C-reactive protein (CRP) |
| Uric acid | creatine phosphokinase (CPK) |

### 2.3.4.2 Urinalysis

A urinalysis will be performed to measure pH, specific gravity, protein (qualitative), glucose (qualitative), ketones (qualitative), bilirubin (qualitative), urobilinogen, occult blood, hemoglobin, and cells. A microscopic examination will be performed, if necessary.

### 2.3.4.3 Pregnancy Test

A serum pregnancy test for human chorionic gonadotropin will be performed on female subjects of childbearing potential at Screening.

A urine dipstick pregnancy test (human chorionic gonadotropin) will be performed on female subjects of childbearing potential at all other study visits as specified in the Time and Events Tables (Table 9 and Table 10).

#### 2.3.5 Adverse Events


An AE is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with study treatment. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The following are not considered to be AEs despite requiring hospitalization:

- , or variations thereof • Pre-existing conditions that, in the opinion of the investigator, did not worsen or progress during study participation
- Routinely scheduled procedures or treatment
- Elective procedures that had been scheduled prior to study participation (i.e., signing of the informed consent form (ICF))

A serious adverse event (SAE) is any untoward medical occurrence that:

- results in death
- is life-threatening (note that this refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe)
- requires hospitalization or prolongation of existing hospitalization
- results in persistent or significant disability/incapacity
- results in a congenital anomaly/birth defect

An SAE may also be any other important medical event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the subject or require intervention to prevent one of the other outcomes listed in the definition above. Examples of such events include intensive treatment in an emergency room or at home for bronchospasm, hyperkalemia, or convulsions that do not result in a formal hospitalization.

Elective hospitalizations scheduled prior to study participation (i.e., signing of the ICF) should not be reported as SAEs.

#### 2.3.6 **Immunogenicity**

antibody (ADA) assessment will be collected as specified in the Time and Events Tables (Table 9 and Table 10) in all enrolled subjects. These samples will be banked and used to investigate and characterize any ADA response over time in the general study population.


#### **Efficacy Assessments**

Higher scores are representative of more severe impairment. Recent data suggest that improvements in the QMG score of 2 to 3 points may be considered clinically meaningful, depending upon disease severity [Barohn, 1998; Katzberg 20147]

Table 2 presents the scoring scale for the 13 individuals he sum of the considered clinically he considered clinically he consi

the sum of the individual scores; range 0 - 39.

If a subject is missing a response for one of the 13 individual QMG items, the subject's corresponding item score from the previously scheduled QMG assessment will be imputed for the missing item score (and the total score calculated using this imputed value and the non-missing item scores). If the item response is also missing from the previously scheduled QMG, the QMG total score will be set to missing for that visit. If the subject is missing responses to more than one of the 13 items, the QMG total score will be set to missing for that visit (note: the LOCF algorithm will still be applied, as appropriate).2.4.2 Myasthenia Gravis Activities of Daily Living Score still be applied, as appropriate).

The MG-ADL is a brief 8-item survey designed to evaluate MG symptom severity. Higher scores are associated with more severe symptoms of MG. The MG-ADL has been shown to correlate with other validated MG outcome measures (e.g., MG-QOL15r), and a 2-point improvement in MG-ADL score is considered clinically meaningful [Wolfe, 1999, Muppidi, 2011].

Table 3 presents the & items with corresponding response scale, each scored on a 0 – 3 point scale (i.e., 0=none, 1=mild, 2=moderate, and 3=severe). The total score is the sum of the 8 individual scores; range 0 - 24.

If a subject is missing a response for one of the 8 individual MG-ADL items, the subject's corresponding item score from the previously scheduled MG-ADL assessment will be imputed for the missing item score (and the total score calculated using this imputed value and the non-missing item scores). If the item response is also unissing from the previously scheduled MG-ADL, the MG-ADL total score will be set to missing for that visit. If the subject is missing responses to more than one of the 8 items, the MG-ADL total score will be set to missing for that visit (note: the LOCF algorithm will still be applied, as appropriate).


#### **Myasthenia Gravis Quality of Life**

myasthenia gravis.

I have limited my social activity because of my myasthenia gravis.

My myasthenia gravis because of my myasthenia gravis.

I have limited my social activity because of my myasthenia gravis.

My myasthenia gravis limits my ability to enjoy hobbies and activities.

I have trouble meeting the needs of my family because of my myasthenia gravis.

I have to make plans around my myasthenia gravis.

My occupational skills and job status have be myasthenia gravis.

I have difficulty speaking.

I have trouble. The MG-QOL15r is a 15-item survey that was designed to assess quality of life in subjects with MG. Higher scores indicate more severe impact of the disease on aspects of the subject's life [Burns, 2010; Burns, 2016].

The following are the 15 questions and the corresponding response scales, each scored on a 0-2 point scale (0=Not much at all, 1=Somewhat, 2=Very Much).

- 11. I am depressed about my myasthenia gravis
- 12. I have trouble walking due to my myasthenia gravis
- 13. I have trouble getting around public places because of my myasthenia gravis.
- 14. I feel overwhelmed by my myasthenia gravis.
- 15. I have trouble performing my personal grooming needs because of myasthenia gravis.

The MG-QOL15r total score is the sum of the 15 individual item scores with a range of 0 - 30.

If a subject is missing a response for one of the 15 individual MG-QOL15r items, the subject's corresponding item score from the previously scheduled MG-QOL15r assessment will be imputed for the missing item score (and the total score calculated using this imputed value and the non-missing item scores). If the item response is also missing from the previously scheduled MG-QOL15r, the MG-QOL15r total score will be set to missing for that visit. If the subject is missing responses to more than one of the 10 items, the MG-QOL15r total score will be set to missing for that visit (note: the LOCF algorithm will still be applied, as appropriate).

### MG Composite

The Chief documents The MG Composite is a 10-item scale that has been used to measure the clinical status of subjects with MG, both in the practice setting and in clinical trials, in order to evaluate treatment response. Higher scores in the MG Composite indicate more severe impairment due to the disease. A 3-point change in this instrument is considered clinically meaningful [Benatar, 2012; Sadjadi, 2012].

> 

Table 4 presents the 10 items with corresponding response scale scores. The total score is the sum of the 10 individual scores; range 0 - 50.

composite items, previously scheduled MG Composite and the non-missing item score (and the total score calculated missing from the previously scheduled MG Composite assessment, the MG Composite total score will be set to missing for that visit. If the subject is missing responses to more than one of the 10 items, the MG Composite total score will be set to missing for that visit (note: the LOCF algorithm will still be applied). a spone ... MG

Ject is missi.

Lotal score will be applied, as applied, as applied, as applied, as applied, as applied and any applied as applied as a support and any applied as a support a

 RA101495-02.201

Table 2: QMG Items and Scoring

| * Circle as appropriate | | | Gra | ade | isio, | | |
|---|---|---|---|---|---|---|---|
| ı | Test Item | Measured value, if applicable | None<br>0 | Mild<br>1 | Moderate 2 | Severe<br>3 | Score<br>(0-3) |
| 1. | Double vision on lateral gaze *right / left / both *glasses removed: Y / N / NA | seconds | ≥61 | 11-60 | on and 1-10 | Spontaneous | |
| 2. | Ptosis<br>(upward gaze) | seconds | ≥61 | 11-60 | 1-10 | Spontaneous | |
| 3. | Facial Muscles | NA | Norma(lid<br>closure | Complete, weak, some resistance | Complete,<br>without<br>resistance | Incomplete | |
| 4. | Swallowing<br>4oz. (½ cup) water | NA ~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~ | Normal | Minimal<br>coughing or<br>throat clearing | Severe<br>coughing/chokin<br>g or nasal<br>regurgitation | Cannot swallow<br>(test not<br>attempted) | |
| 5. | Speech after counting aloud from #1 to 50 | Number | None at<br>#50 | Dysarthria at<br>#30-49 | Dysarthria at<br>#10-29 | Dysarthria at<br>9 | |
| 6. | Right arm outstretched (90°, sitting, away from back of chair) | Seconds | 240 | 90-239 | 10-89 | 0-9 | |
| 7. | Left arm outstretched<br>(90°, sitting, away from<br>back of chair) | seconds | 240 | 90-239 | 10-89 | 0-9 | |


### Statistical Analysis Plan

| 8. | Forced vital capacity FVC % predicted [%p] FVC [L] | Best of 3-5 attempts%pFVC [L] Normal Range used: NHANES III | ≥80% | 65-79% | 50-64% | si <sup>01</sup> <50% |
|---|---|---|---|---|---|---|
| 9. | Right hand grip<br>Men<br>Women | *Setting: 2 3 | ≥45<br>≥30 | 15-44<br>10-29 | 5-14<br>5-9 | 0-4<br>0-4 |
| 10. | Left hand grip<br>Men<br>Women | *Setting: 2 3 | ≥35<br>≥25 | 15-34<br>10-24 | 5-14<br>5-9 | 0-4<br>0-4 |
| 11. | Head, lifted<br>(45°, supine) | seconds | 120 | 30-119 | 1-29 | 0 |
| 12. | Right leg outstretched (45°, supine) | seconds | 100 <sup>C</sup> 21/1/1 | 31-99 | 1-30 | 0 |
| 13. | Left leg outstretched (45°, supine) | seconds | 100 | 31-99 | 1-30 | 0 |


**Table 3: MG-ADL Items and Scoring** 

| Grade | 0 | 1 | 2 | 3 | Score |
|---|---|---|---|---|---|
| Talking | Normal | Intermittent<br>slurring of nasal<br>speech | Constant slurring or nasal, but can be understood | Difficult to understand speech | ijonsim |
| Chewing | Normal | Fatigue with solid food | Fatigue with soft food | Gastric tube | |
| Swallowing | Normal | Rare episode of choking | Frequent choking necessitating changes in diet | Gastric tube | |
| Breathing | Normal | Shortness of breath with exertion | Shortness of breath at rest | Ventilator<br>dependence | |
| Impairment of ability<br>to brush teeth or<br>comb hair | None | Extra effort, but no rest periods needed | Rest periods<br>needed | Cannot do one of these functions | |
| Impairment of ability to arise from a chair | None | Mild, sometimes<br>uses arms | Moderate, always<br>uses arms | Severe, requires assistance | |
| Double vision | None | Occurs, but not daily | Daily, but not constant | Constant | |
| Eyelid droop | None | Occurs, but not<br>daily | Daily, but not constant | Constant | |
| not be used to | | | | | |


Table 4: MG-Composite Assessments and Scoring

| | | Item | Seconds,<br>if applicable | | | Ś | ons | Score |
|---|---|---|---|---|---|---|---|---|
| Transcribe from QMG | 1. | Ptosis<br>upward ease, seconds<br>(physician examination) | seconds | >45<br>seconds<br>=0 | 11-45<br>=1 | 1-10-1 | Immediate<br>=3 | |
| | 2. | Double vision<br>on lateral gaze<br>left/right/both, seconds<br>(physical examination) | seconds | >45<br>seconds<br>=0 | 11-45<br>=1 | 1-10<br>=3 | Immediate<br>=4 | |
| Transcri | 3. | Eye closure<br>(physician examination) | NA | Normal<br>=0 | Mild weakness<br>(can be forced<br>open with<br>effort)<br>=0 | Moderate weakness (can be forced open easily) =1 | Severe weakness (unable to keep eye closed) =2 | |
| MG-ADL | 4. | Talking<br>(patient history) | NA | Normal<br>=0 | Intermittent slurring or nasal speech =2 | Constant slurring or nasal but can be understood = 4 | Difficult to<br>understand<br>speech<br>=6 | |
| Transcribe from MG-ADL | 5. | Chewing<br>(patient history) | NA and | Normal<br>=0 | Fatigue with solid food =2 | Fatigue with soft food =4 | Gastric tube<br>=6 | |
| Transcri | 6. | Swallowing<br>(patient history) | NA NA | Normal<br>=0 | Rare episode of choking or trouble swallowing =2 | Frequent<br>trouble<br>swallowing<br>=5 | Gastric Tube<br>=6 | |


### Statistical Analysis Plan

| | | | | | | ~ ~ ~ |
|---|---|---|---|---|---|---|
| 7 | 7. Breathing thought to be caused by MG (patient history) | NA | Normal<br>=0 | Shortness of breath with exertion =2 | Shortness of<br>breath at rest<br>=4 | Ventilator<br>dependence<br>=9 |
| 8 | Neck flexion or extension (weakest) (physician examination) | NA | Normal<br>=0 | Mild weakness<br>=1 | Moderate<br>weakness | Severe<br>weakness<br>=4 |
| 9 | 9. Shoulder abduction (physician examination) | NA | Normal<br>=0 | Mild weakness<br>=2 | Moderate<br>weakness<br>=4 | Severe<br>weakness<br>=5 |
| 10 | Hip Flexion (physician examination) | NA | Normal<br>=0 | Mild weakness | Moderate<br>weakness<br>=4 | Severe<br>weakness<br>=5 |


#### 2.5 Pharmacokinetic Assessments

| 2.5 Pharmacokinetic Assessments | | | |
|---|---|---|---|
| The following are the Pharmacokinetic (PK) endpoints: | | | |
| The following are the Pharmacokinetic (PK) endpoints: Plasma concentrations of RA101495 and its major metabolites Maximum plasma concentration (C <sub>max</sub> ) on Day 1 Time corresponding to C <sub>max</sub> (t <sub>max</sub> ) on Day 1 Ratio of parent to metabolites (i.e., 2 metabolites). Table 5 and Table 6 present the schedule of PK blood samples for the Main Portion | | | |
| Table 5 and Table 6 pri and Extension Portion Table 5: Main Portion: P | , respectively. | • | he Main Portion |
| Day 1 | Day 84 | At sites where rescue therapy is administered | at sites where rescue therapy is NOT |
| · | | At sites where rescue<br>therapy is administered<br>locally | At sites where rescue<br>therapy is NOT<br>administered locally |
| predose | predose | At sites where rescue therapy is administered locally Within 1 hour before | At sites where rescue therapy is NOT administered locally Prior to administration of |
| predose<br>(within 1 hour before first | predose<br>(any time prior to Day 84 | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue |
| predose<br>(within 1 hour before first<br>dose of study drug) | predose<br>(any time prior to Day 84<br>study drug administration) | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy | At sites where rescue therapy is NOT administered locally Prior to administration of |
| predose<br>(within 1 hour before first | predose<br>(any time prior to Day 84 | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy |
| predose (within 1 hour before first dose of study drug) 1 hour postdose | predose (any time prior to Day 84 study drug administration) 1 hour postdose | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy For PLEX only PK will be | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy After administration of the |
| predose (within 1 hour before first dose of study drug) 1 hour postdose (± 30 minutes) 3 hours postdose | predose (any time prior to Day 84 study drug administration) 1 hour postdose | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy For PLEX only: PK will be measured in the exchanged plasma Within 1 hour after | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy After administration of the last course of rescue |
| predose<br>(within 1 hour before first<br>dose of study drug)<br>1 hour postdose<br>(± 30 minutes) | predose (any time prior to Day 84 study drug administration) 1 hour postdose | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy For PLEX only: PK will be measured in the exchanged plasma Within 1 hour after administration of rescue | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy After administration of the last course of rescue |
| predose (within 1 hour before first dose of study drug) 1 hour postdose (± 30 minutes) 3 hours postdose (± 30 minutes) | predose (any time prior to Day 84 study drug administration) 1 hour postdose | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy For PLEX only: PK will be measured in the exchanged plasma Within 1 hour after | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy After administration of the last course of rescue |
| predose (within 1 hour before first dose of study drug) 1 hour postdose (± 30 minutes) 3 hours postdose | predose (any time prior to Day 84 study drug administration) 1 hour postdose | At sites where rescue therapy is administered locally Within 1 hour before administration of rescue therapy For PLEX only: PK will be measured in the exchanged plasma Within 1 hour after administration of rescue | At sites where rescue therapy is NOT administered locally Prior to administration of the first course of rescue therapy After administration of the last course of rescue |

Table 6: Extension Portion: Pharmacokinetic Schedule of Assessments

| During Resc | Week E36 | |
|---|---|---|
| At sites where rescue therapy is administered locally | At sites where rescue therapy is NOT administered locally | (see Study Protocol Appendix 2) |
| Within 1 hour before administration | Prior to administration of the first | predose (within 1 hour before first |
| of rescue therapy | course of rescue therapy | dose of study drug) |
| For PLEX only: PK will be measured | After administration of the last | 1 hour postdose (± 30 minutes) |
| in the exchanged plasma | course of rescue therapy | |
| Within 1 hour after administration of | | 3 hours postdose (± 30 minutes) |
| rescue therapy | | |
| C.O | | 6 hours postdose (± 90 minutes) |

On all other study visit days, a single PK sample will be collected prior to administration of study drug. Plasma concentrations of RA101495 and its metabolites will be measured and reported in all subjects receiving RA101495. All samples will be sent to a central laboratory for analysis. Detailed instructions regarding PK sample collection, processing, and shipping will be provided to sites.

#### 2.6 **Pharmacodynamic Assessments**

The following are the Pharmacodynamic assessments:


RA101495-02.201

Statistical Analysis Plan

- Sheep red blood cell (sRBC) lysis assay for evaluation of classical complement pathway activation
- C5 levels.

Table 7 and Table 8 present the schedule of Pharmacodynamic (PD) blood samples for the Main Portion and Extension Portion, respectively.

Table 7: Main Portion: Pharmacodynamic Schedule of Assessments

| | | During Reso | rue Therapy* |
|---|---|---|---|
| Day 1 | Day 84 | At sites where rescue<br>therapy is NOT<br>administered locally | |
| predose | predose | Within 1 hour before | Prior to administration of |
| (within 1 hour before first | (any time prior to Day 84 | administration of rescue | the first course of rescue |
| dose of study drug) | study drug administration) | therapy | therapy |
| 1 hour postdose | 1 hour postdose | | 40 |
| (± 30 minutes) | (± 30 minutes) | | |
| 3 hours postdose | | Within 1 hour after | After administration of the |
| (± 30 minutes) | | administration of rescue | last course of rescue |
| | | therapy | therapy |
| 6 hours postdose | | inerapy :: Callott | |
| (± 90 minutes) | | | |

Table 8: Extension Portion: Pharmacodynamic Schedule of Assessments

| During Resc<br>(ONLY throug | Week E36 | |
|---|---|---|
| At sites where rescue therapy is administered locally | At sites where rescue therapy is NOT administered locally | (see Study Protocol Appendix 2) |
| Within 1 hour before administration | Prior to administration of the first | predose (within 1 hour before first |
| of rescue therapy | course of rescue therapy | dose of study drug) |
| For PLEX only: PK will be measured | After administration of the last | 1 hour postdose (± 30 minutes) |
| in the exchanged plasma | course of rescue therapy | |
| Within 1 hour after administration of | N. C. | 3 hours postdose (± 30 minutes) |
| rescue therapy | 20° | |
| | 11. | 6 hours postdose (± 90 minutes) |

# 2.7 Rescue Therapy

Subjects are expected to remain on stable doses of standard of care therapy for gMG throughout the Main Portion of the study and through the Day E84 visit of the Extension Portion, including pyridostigmine, corticosteroids, or immunosuppressive drugs. If, in the opinion of the investigator, escalation of gMG therapy (i.e., 'rescue therapy') becomes necessary due to deterioration of a subject's clinical status, the subject may receive immunoglobulin or plasma exchange treatment. If such rescue therapy becomes necessary, the choice of immunoglobulin vs. plasma exchange, as well as the frequency and duration of such therapy, will be determined by the investigator. Escalation of doses of pyridostigmine, corticosteroids, or immunosuppressive drugs for rescue is not permitted.

A Rescue Therapy Visit should be performed prior to initiation of rescue therapy (see Table 9 and Table 10 for a list of applicable study procedures).


RA101495-02.201

Statistical Analysis Plan

e 9) and the probability of the

 RA101495-02.201

### Statistical Analysis Plan

**Table 9: Main Portion: Time and Events Table** 

| Study Procedure | Screening<br>Days -28 to -1 | Day 1 | Day 8<br>(± 2 days) | Day 15<br>(± 2 days) | Day 29 (± 2 days) | Day 57 (± 7 days) | End of Study <sup>a</sup> Day 84 (± 2 days) | Safety<br>Follow-up Call<br>(last dose + 40d) | Rescue Therapy Visit <sup>b</sup> (if applicable) |
|---|---|---|---|---|---|---|---|---|---|
| Informed consent <sup>c</sup> | X | | | | | | . ( | | |
| Review eligibility and randomization <sup>c</sup> | X | | | | | | 5 | | |
| Medical history <sup>d</sup> and demographics | X | | | | | | ,01 | | |
| Height <sup>e</sup> and weight | X | | | | X | | X | | |
| Prior and concomitant medications <sup>f</sup> | X | X | X | X | X | X | √ X | | X |
| Safety | | | | | | | | | |
| Physical examination <sup>g</sup> | X | X | X | X | X | X | X | | X |
| Vital signs <sup>h</sup> | X | X | X | X | X | X | X | | X |
| 12-Lead electrocardiogram | X | | | | | | X | | X |
| Neisseria meningitidis vaccinationi | X | | | | | illo | | | |
| Hematology/Chemistry <sup>j</sup> | X | X | X | X | X | COX | X | | X |
| Coagulation <sup>k</sup> | X | X | X | X | $\int X \propto 0$ | X | X | | X |
| Urinalysis | X | X | X | X | $X \times X$ | X | X | | X |
| Pregnancy test <sup>1</sup> | X | X | | | 100 | | X | | |
| Adverse events <sup>m</sup> | | X | X | X | X | X | X | X <sup>m</sup> | X |
| Anti-drug antibody | X | | | × × × | X | | X | | X |
| Efficacy | | | ( | , , , , , , , | | | | | |
| QMG Test/Score <sup>n</sup> | X | X | X | X | X | X | X | | X |
| MG-ADL | | X | X | ΟX | X | X | X | | X |
| MG-QOL15r | | X | ₹ | > X | X | X | X | | X |
| MG Composite | | X | X | X | X | X | X | | X |
| Pharmacokinetic/Pharmacodynamic | | | il. | | | | | | |
| RA101495 plasma PK° | | Xº | X | X | X | X | Xº | | Xº |
| Pharmacodynamic analysis <sup>o</sup> | | X° \ | X | X | X | X | Xº | | Xº |
| Exploratory | | ar | , | | | | | | |
| Additional biomarker samples <sup>p</sup> | | X | X | X | X | X | X | | |
| Pharmacogenomic analysis (optional) | X | 00, | | | | | | | |
| Study Drug | ,, | 64 | | | | | | | |
| RA101495 or placebo administration <sup>q</sup> | ,0<br>S, | X | X | X | X | X | X | | Xq |

See footnotes on following page.


#### RA101495-02.201

#### Statistical Analysis Plan

- 1-a. If a subject prematurely discontinues study drug at any time prior to completion of the Day 84 visit during the Treatment Period, the subject should return to clinic for an End of Study Visit.
- 1-b. For subjects who require rescue therapy (see Protocol Section 10.1.3.1), a Rescue Therapy Visit should be conducted prior to the initiation of rescue therapy. If the Rescue Therapy Visit coincides with a regularly scheduled study visit, then overlapping study procedures do not need to be duplicated.
- 1-c. Procedures performed as SOC during the Screening Period may be used to determine eligibility. Informed consent must be obtained prior to performing any study-specific procedures that are not SOC.
- 1-d. Screening includes disease history with diagnosis of gMG by the MGFA criteria (Class II-IVa), serology for AChR autoantibodies
- 1-e. Height will be measured only at Screening.
- 1-f. All prescriptions and over-the-counter medications taken during the 30 days prior to baseline (i.e., Day 1) through the last study visit will be documented. NOTE: A complete history of medications taken for the treatment of gMG will be collected.
- 1-g. A full physical examination will be performed on all subjects at Screening. On all other study visit days, the physical examination will be symptom-directed.
- 1-h. The vital signs assessment will include measurement of HR, body temperature, and blood pressure in the sitting position.
- 1-i. All subjects must have documentation of prior *Neisseria meningitidis* vaccination (and booster, if appropriate) prior to study entry. If the subject has not been vaccinated, he/she must be vaccinated with a quadrivalent meningococcal vaccine at least 14 days prior to the first dose of study drug on Day 1 and should have a booster vaccination as indicated by SOC. Subjects should bring their patient safety card to every study visit. If the subject does not bring their card with them they will be given a new one.
- 1-j. All laboratory samples should be obtained prior to administration of study drug at applicable visits unless otherwise noted for PK, PD, and biomarker samples.
- 1-k. Coagulation tests should be performed only in subjects who are receiving anticoagulant therapy.
- 1-l. For all female subjects of childbearing potential, a negative serum pregnancy test must be documented at Screening. All other pregnancy tests will be performed via urine.
- 1-m. All AEs and SAEs should be monitored until resolution or stabilization. SAEs that occur within 40 days after the last dose of study drug should be reported using the procedures outlined in the protocol. Sites will call subjects 40 days after their last dose to gather information on ongoing AEs and report any new SAEs since the last study visit. This Safety Follow-up Call will only be required for subjects who choose not to receive RA101495 in the Extension Portion.
- 1-n. The assessment of QMG should be performed at approximately the same time of day (preferably in the morning) and administered by the same well-trained evaluator (e.g., neurologist, physical therapist, or other study staff) at each visit throughout the study. If a subject is receiving a cholinesterase inhibitor, the dose must be withheld for at least 10 hours prior to the OMG test.

1-o. Blood samples for PK and PD analysis will be obtained at the following time points:

| | 4 | During Reso | cue Therapy |
|---|---|---|---|
| Day 1 | Day 84 | At sites where rescue therapy is administered locally | At sites where rescue therapy is NOT administered locally |
| predose (within 1 hour before first dose of | predose (any time prior to Day 84 study drug | Within 1 hour before administration of rescue | Prior to administration of the first course of |
| study drug) | administration) | therapy | rescue therapy |
| 1 hour postdose (± 30 minutes) | 1 hour postdose (± 30 minutes) | For PLEX only: PK will be measured in the | After administration of the last course of |
| | *O | exchanged plasma | rescue therapy |
| 3 hours postdose (± 30 minutes) | 7.00 | Within 1 hour after administration of rescue | |
| | 20 | therapy | |
| 6 hours postdose (± 90 minutes) | Ī | | |

On all other study visit days, PK/PD samples should be collected prior to administration of study drug.

- 1-p. Blood samples for biomarker testing will be obtained prior to administration of study drug (within 1 hour of dosing) and at 6 hours postdose (± 90 minutes) on Day 1. On all other study visit days, biomarkers samples should be collected prior to administration of study drug.
- 1-q. Dosing on study visit days should be held until QMG scoring, PK, and PD sample blood collection has been completed. On days when rescue therapy is concurrently administered, study drug dosing should be held until after administration of rescue therapy and PK/PD sampling.


Table 10: **Extension Portion: Time and Events Table** 

| Study Procedure | Day E1 <sup>a</sup> (Day 84) | Day E8<br>(± 2 days) | Day E15<br>(± 2 days) | Day E29<br>(± 2 days) | Day E57<br>(± 7 days) | Day E84 (± 7 days) | Rescue<br>Therapy Visit <sup>b</sup><br>(if applicable) | ionsol | Final Study<br>Visit <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | | | | | | 25 | | |
| Review eligibility and randomization | X | | | | | | To | | |
| Weight | X | | | X | | X | , 0, | | X |
| Prior and concomitant medications | X | X | X | X | X | X | (X) | | X |
| Safety | | | | | | | 70. | | |
| Physical examination (symptom directed) | X | X | X | X | X | X | X | | X |
| Vital signs <sup>d</sup> | X | X | X | X | X | X | O X | | X |
| 12-Lead electrocardiogram | | | | | | X <sub>1</sub> O <sup>1</sup> | X | S | X |
| Neisseria meningitidis vaccinatione | SOCe | | | | | CO. | | Dud | |
| Hematology/Chemistry <sup>f</sup> | X | X | X | X | X | All X | X | y F | X |
| Coagulation <sup>g</sup> | X | X | X | X | OX o | X | X | Please refer to | X |
| Urinalysis | X | X | X | X | $O^{X}$ | X | X | ase | X |
| Pregnancy test <sup>h</sup> | X | | | | 10,0 | X | | ref<br>ol | X |
| Adverse eventsi | X | X | X | X.V | ΛŌX | X | X | Apj | X |
| Anti-drug antibody | X | | | CX C | | X | X | per to | X |
| Efficacy | | | | 10 ×10 | , | | | Please refer to Study Protocol Appendix 2 | |
| QMG Test/Score <sup>j</sup> | X | X | X | ) X) | X | X | X | x 2 | X |
| MG-ADL | X | X | X <sub>2</sub> V | -OX | X | X | X | | X |
| MG-QOL15r | X | X | X | X | X | X | X | | X |
| MG Composite | X | X | X | X | X | X | X | | X |
| Pharmacokinetic/Pharmacodynamic | | | -0/ | | | | | | |
| RA101495 plasma PK <sup>k</sup> | $X^k$ | X | X | X | X | X | $X^k$ | | X |
| Pharmacodynamic analysis <sup>k</sup> | $X^k$ | X | (3) X | X | X | X | $X^k$ | | X |
| Exploratory | | × 2 | <i>Y</i> | | | | | | |
| Additional biomarker samples <sup>1</sup> | $X^{l}$ | X | X | X | X | X | | | X |
| Study Drug | | .09 | | | | | | | |
| RA101495 administration <sup>m</sup> | X | X | X | X | X | X | X <sup>m</sup> | | X |

See footnotes on following page.


#### RA101495-02.201

#### Statistical Analysis Plan

- 2-a. For subjects that decide and are eligible to continue in the Extension Portion, the Day 84 visit from the Main Portion will serve as the Day E1 visit and will also include review of eligibility to continue, treatment group assignment (see Protocol Section 8.3), signing of an informed consent for the Extension Portion, and an additional biomarker blood sample.
- 2-b. For subjects who require rescue therapy (see Protocol Section 10.1.3.1), a Rescue Therapy Visit should be conducted prior to the initiation of rescue therapy. If the Rescue Therapy Visit coincides with a regularly scheduled study visit, then overlapping study procedures do not need to be duplicated.
- 2-c. If a subject discontinues study drug treatment at any time during the Extension Period, the subject should return to clinic for a Final Study Visit.
- 2-d. The vital signs assessment will include measurement of HR, body temperature, and blood pressure in the sitting position.
- 2-e. During the Extension Portion, all subjects should have *Neisseria meningitidis* booster vaccinations as indicated by SOC. Subjects should bring their patient safety card to every study visit. If the subject does not bring their card with them they will be given a new one.
- 2-f. All laboratory samples should be obtained prior to administration of study drug at applicable visits unless otherwise noted for PK, PD, and biomarker samples.
- 2-g. Coagulation tests should be performed only in subjects who are receiving anticoagulant therapy.
- 2-h. Urine pregnancy tests will be conducted in female subjects of childbearing potential.
- 2-i. All AEs and SAEs should be monitored until resolution or stabilization. SAEs that occur within 40 days after the last dose of study drug should be reported using the procedures outlined in the protocol.
- 2-j. The assessment of QMG should be performed at approximately the same time of day (preferably in the morning) and administered by the same well-trained evaluator (e.g., neurologist, physical therapist, or other study staff) at each visit throughout the study. If a subject is receiving a cholinesterase inhibitor, the dose must be withheld for at least 10 hours prior to the QMG test.

2-k. Blood samples for PK and PD analysis will be obtained at the following time points:

| Day E1 | During Rescue Therapy | |
|---|---|---|
| (Day 84 from the Main Portion) | At sites where rescue therapy is administered locally | At sites where rescue therapy is NOT administered locally |
| predose (any time prior to Day 84 study | Within 1 hour before administration of | Prior to administration of the first course |
| drug administration) | rescue therapy | of rescue therapy |
| 1 hour postdose (± 30 minutes) | For PLEX only: PK will be measured in | After administration of the last course of |
| | the exchanged plasma | rescue therapy |
| | Within 1 hour after administration of | |
| | rescue therapy | |
| | · 4 | |

On all other study visit days, PK/PD samples should be collected prior to administration of study drug.

- 2-1. Biomarkers samples should be collected prior to administration of study drug.
  - NOTE: For those subjects that consent to the Extension Portion an additional blood sample for biomarker testing will be taken at 6 hours postdose (± 90 minutes) on Day 84.
- 2-m. Dosing on study visit days should be held until QMG scoring, PK, and PD sample blood collection has been completed. On days when rescue therapy is concurrently administered, study drug dosing should be held until after administration of rescue therapy and PK/PD sampling.


#### 3 STATISTICAL METHODS

#### 3.1 General Methods

#### 3.1.1 Computing Environment

All statistical analyses will be performed using SAS® Version 9.1.3 or higher for Windows.

### 3.1.2 Reporting of Numerical Values

30ns of variations thereof. All clinical study data will be presented in subject data listings. Descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) will be calculated by treatment group for continuous variables. Confidence intervals will be provided where appropriate. For continuous endpoints, the confidence interval for the mean will be based on the t-distribution (e.g., CLM in the SAS Proc Means procedure).

Frequencies and percentages will be presented by treatment group for categorical and ordinal variables. If there are missing values, the number of missing values will be presented, but without a percentage and the number of non-missing values used as the denominator.

Means, medians, standard deviations, and confidence intervals will be reported to one decimal place more than the data reported on the CRF or by the laboratory/vendor. Minimum and maximum will be reported to the same number of decimal places displayed on the CRF or by the laboratory/vendor. P-values will be reported to 4 decimal places.

### 3.1.3 Baseline Value and Change from Baseline

Unless otherwise specified, for the Main Portion analyses, the baseline value is defined as the most recent non-missing value obtained prior to the subject receiving the first dose of study drug. For most endpoints this will be the Day 1 visit assessment.

For analyses which include the Extension Portion, some analyses may utilize a "baseline" defined as the value obtained prior to receiving the first administration of RA101495 (i.e., first dose of active treatment). For subjects who received RA101495 same, the most recent non-missing subjects received placebo in the Main Portion, the value obtained prior to receiving the first administration of RA101495 will generally occur on the Day E1 (Day 84) visit, and will be the baseline value.

The cases where baseline is defined as the value receiving the first administration. during the Main Portion, the baseline remains the same, the most recent non-missing value obtained prior to the subject receiving the first dose of study drug. For subjects


#### 3.2 Handling of Missing Values

#### 3.2.1 Efficacy Endpoints: Main Portion

The primary method for handling missing data in the efficacy analyses will be last observation carried forward (LOCF). For the LOCF algorithm, if a patient is missing a value, the closest non-missing endpoint value prior to the missing value will be imputed for the missing value (note: this includes the baseline value and values from unscheduled visits).

Variations thereof. Additionally, if a subject receives rescue therapy (see Section 2.7), efficacy endpoints occurring after rescue therapy will be censored and imputed using the LOCF method. The LOCF method is such that the closest non-missing endpoint value prior to the initiation of rescue therapy will be imputed, (note: this includes the baseline value and values from unscheduled visits).

For selected efficacy endpoints, observed case analyses will be presented as a sensitivity analysis.

Observed Case Method: analyses censoring observations post-rescue therapy medication. Observations occurring post-rescue therapy will be censored and not imputed. Otherwise, missing values will not be imputed. Note that the imputation of individual efficacy assessment items to create a total score, as discussed in Section 2.4 will still be applied in the Observed Case Method.

### 3.2.2 Efficacy Endpoints: Extension Portion

For analyses which involve the Extension Portion (i.e., analyses of the Extension Period data or analyses combining the Main and Extension Periods), the following methods will be applied to the Extension Portion efficacy analyses:

LOCF method in Extension Period:

If a subject is missing values for a scheduled assessment the subject's previous non-missing value will be imputed (note: this includes the baseline value and values from unscheduled visits).

### Handling of Values Post-Rescue Medication Use:

If the subject was in one of the active treatment groups in the Main Portion of

If the subject the study: If the subject had received rescue medication in the Main Portion of the study (see Section 2.7), then the subject will continue to have postrescue medication observations censored and imputed using LOCF method in the Extension Period.

If the subject had not received rescue medication in the Main Portion of the study but receives rescue medication in the Extension Period, the post-rescue medication observations will be censored and imputed


RA101495-02.201

Statistical Analysis Plan

via LOCF method (i.e., using the methodology described in Section 3.2.1).

If the subject was in the placebo treatment group in the Main Portion of the study:

It the subject had received rescue medication in the Main Portion of the study (see Section 2.7), the subject will stop having the post-rescue medication observations censored after, but not including, the Day 840 visit (i.e., LOCF in the Main Portion will not carry over interest Extension Portion).

If the subject receives rescue medication in the Extension Period, the post-rescue medication observations will be censored and imputed via LOCF method (i.e., using the methodology described in Section 3.2.1).

Observed Case Method in Extension Portion:

Missing values will not be imputed, and analyses will be performed on the observed cases (with the exception of observations occurring post-rescue medication use). Note that the imputation of individual efficacy assessment items to create a total score, as discussed in Section 2.4, will still be applied in the Observed Case Method.

# Handling of Values Post-Rescue Medication Use:

If the subject was in one of the active treatment groups in the Main Portion of the study:

• If the subject had received rescue medication in the Main Portion of the study (see Section 2.7), then the subject will continue to have postrescue medication observations censored in the Extension Period.

If the subject had not received rescue medication in the Main Portion of the study but receives rescue medication in the Extension Period, the post-rescue medication observations will be censored.

If the subject was in the placebo treatment group in the Main Portion of the study:

If the subject had received rescue medication in the Main Portion of the study (see Section 2.7), the subject will stop having the post-rescue medication observations censored after, but not including, the Day 84 visit (i.e., the censoring of observations in the Main Portion will not carry over into the Extension Portion).


RA101495-02.201

Statistical Analysis Plan

If the subject receives rescue medication in the Extension Period, the post-rescue medication observations will be censored.

J.3 Analysis Populations

Analysis populations are identical, duplicate results may not be presented for the identical populations.

3.3.1 Intention-to-Treat Population

The Intention-to-Treat (ITT) Population opulation analyses will be 1

#### 3.3.2 Modified ITT Population

The modified ITT (mITT) Population will include all subjects in the ITT Population who have received at least 1 dose of study drug, mITT population analyses will be based on the randomized treatment.

#### 3.3.3 Per Protocol Population

The Per Protocol Population will include all subjects in the mITT Population who have completed the 12-week Treatment Period and have no major protocol violations during the 12-week Treatment Period.

If, in the Main Portion of the study, a patient received multiple doses of different study drug levels (i.e., placebo, 0.1 mg/kg, and 0.3 mg/kg), the patient will be assigned to the dose group which they received at the highest frequency within the Main Portion of the study.

Similarly, if in the Extension Portion of the study, a patient received multiple doses of different study drug levels (i.e., 0.1 mg/kg, and 0.3 mg/kg), the patient will be assigned to the dose group which they received at the highest frequency within the Extension Portion of the study.

#### 3.3.4 **Safety Population**

The Safety Population will include all subjects who have received at least 1 dose of study drug (i.e., mITT Population), with subjects to be analyzed based on the actual treatment received.


RA101495-02.201

Statistical Analysis Plan

If, in the Main Portion of the study, a patient received multiple doses of different study drug levels (i.e., placebo, 0.1 mg/kg, and 0.3 mg/kg), the patient will be assigned to the dose group which they received at the highest frequency within the

Joseph Green Study.

J.3.5 RA101495 Safety Population

The RA101495 Safety Population will include all subjects who are assigned to an active treatment group in the Main Portion of the study in the Safety Population or received at least 1 dose of RA10495 in the Extension Portion (i.e., this power would not include subjects who, in the Safety Population. We blacebo group in the Main Portion and dropped (A101495).

The Main Portion and dropped (A101495).

study drug levels (i.e., placebo, 0.1 mg/kg, and 0.3 mg/kg), the patient will be assigned to the dose group which they received at the highest frequency within the Main Portion of the study.

Similarly, if in the Extension Portion of the study, a patient received multiple doses of different study drug levels (i.e., 0.1 mg/kg, and 0.3 mg/kg), the patient will be assigned to the dose group which they received at the highest frequency within the Extension Portion of the study.

#### 3.3.6 Pharmacokinetic Population

The PK Population will include all subjects in mITT Population who have at least 1 evaluable PK assessment, All PK analyses will be performed using this population.

## 3.3.7 Pharmacodynamic Population

The PD Population will include all subjects in mITT Population who have at least 1 evaluable PD assessment. All PD analyses will be performed using this population.

### **Combining RA101495 Data Across Study Portions**

For many of the efficacy and safety endpoints, the data from the Main Portion and the Extension Portion will be combined and summarized. Specifically, the Main Portion data for subjects in the 0.1 mg/kg dose group will be combined with the Extension Portion data for subjects in the placebo—0.1 mg/kg group (i.e., subjects in the placebo group for the Main Portion who receive 0.1 mg/kg in the Extension Portion). For the efficacy and safety data, the schedule of assessments between the Main Portion and Extension Portion are such that the scheduled assessments match up as is indicated by the "E1", "E8",..., "E84" naming convention used for the Extension Portion visit


RA101495-02.201

Statistical Analysis Plan

dates (see Table 10). The same combining of data procedure will be applied to the 0.3 mg/kg dose group as well.

Efficacy Endpoints

The following are the primary and secondary efficacy endpoints. For these endpoints baseline will be based on Day 1 value.

3.5.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the change of QMG score.

### 3.5.2 Secondary Efficacy Endpoints

The key secondary efficacy endpoint is change from baseline to Week 12 in the MG-ADL scale.

Additional secondary efficacy endpoints are:

- Change from baseline to Week 12 in the MG-ADL scale
- Minimal symptom expression at Week 12, defined as an MG-ADL scale score of 0 or 1
- Change from baseline to Week 12 in the MG-Quality of Life 15r (MG-QOL15r) survey
- Change from baseline to Week 12 in the MG Composite
- $A \ge 3$ -point reduction in QMG score at Week 12
- Requiring rescue therapy over the 12-week Treatment Period.

#### 3.6 Pharmacodynamic Endpoints

The PD assessments are:

- Sheep red blood cell (sRBC) lysis assay for evaluation of classical complement pathway activation
- C5 levels

### **Exploratory Endpoints**

The following exploratory endpoints will also be examined during the study:

- Responder analysis for changes in QMG, MG-ADL, MG-QOL, and MG-Composite Scores from baseline to Week 12.
- Functional sub-scores of the QMG, MG-ADL, MG-QOL, and MG-Composite scores


o Items for the functional scales are defined in Table 11. The functional subscore for a subject is defined as the total score of the corresponding items (or the value of the item if it is a single score).

| <b>Table</b> | 11. | Fur | etion | al S | hih_ | Scares |
|--------------|-----|------|---------|------|---------|--------|
| Lame | 11. | ı uı | ICLIVII | | , u 1/- | DUDIES |

| | | Scales | | |
|-------------|-----------|--------|--------|--------------|
| Function | QMG | MG ADL | QOL | MG Composite |
| Ocular | 1-3 | 7-8 | 2 | 1-3 |
| Bulbar | 4-5 | 1-3 | 3, 9 | 4-6 |
| Respiratory | 8 | 4 | | 7 60 |
| Limb/Axial | 6-7, 9-13 | 5-6 | 12, 15 | 8-10 |

If an item response has a missing value, the methods defined in Section 2.4 for imputing missing values will be used. Specifically, if a subject is missing a response for one of the items, the subject's corresponding item score from the previously scheduled assessment will be imputed for the missing item score (and the total score calculated using this imputed value and the non-missing item scores). If the item response is also missing from the previously scheduled assessment, the corresponding function sub-score will be set to missing.

- Mechanistic biomarkers [e.g., MG pathophysiology, complement fixation, complement function, complement pathway proteins, autoantibody characterization (titer and immunoglobulin class) and inflammation]
- Pharmacogenomic analyses (optional)

# 3.8 Patient Disposition and Evaluability

## 3.8.1 Patient Disposition

A disposition of all randomized subjects will be provided. This will include the number and percentage of subjects evaluated for each of the analysis populations (Section 3.3), which will be presented by treatment group and overall. Percentages will be based on the number of subjects in the ITT population in the respective treatment group and overall unless otherwise specified.

The number of subjects completing the Main Portion, entering the Extension Portion, completing study Visit Day E84 (i.e., Day 84 of the Extension Portion), discontinuing from the study, and the primary reason for discontinuation will also be summarized.

#### 3.8.2 Protocol Deviations

A listing of protocol deviations will be presented by treatment group.


#### 3.9 Demographics and Baseline Characteristics

#### 3.9.1 Demographics

Subject demographics and baseline characteristics will be summarized by treatment group and overall for the ITT, mITT, Safety, and PP Populations.

, or variations thereof. Descriptive statistics will be provided for age, height, weight, and body mass index (BMI, calculated as weight in kilograms divided by height in meters squared). Frequencies and percentages will be tabulated for sex, race, and ethnicity. Age will also be summarized by <65, 65-<75, and  $\ge 75$ .

Age will be calculated as (informed consent date – date of birth + 1)/365.25, truncated and displayed as years. BMI will be calculated as weight (kg)/height<sup>2</sup> (m<sup>2</sup>), using the weight and height measurements obtained at screening.

Baseline and Screening QMG scores will be summarized. Additionally, for Screening QMG, the number and percentage of patients with scores  $\leq 17 / \geq 18$  will be presented. Baseline MG-ADL will also be summarized.

Note: If the day and month are missing for date of birth, impute January 1st, if only the day is missing impute the 1<sup>st</sup>.

Two-sided p-values will be calculated comparing the similarity of the distribution of the demographics and baseline characteristics across the treatment groups. For the continuous endpoints, the p-value from the overall F-test from an analysis of variance (ANOVA) with treatment group as the factor will be presented. (Note: the set of continuous endpoints are: age, weight, BMI, Screening QMG score, Baseline QMG Score, Baseline ADL score). For categorical variables the p-value from the 3×2 Fisher's exact test will be presented, with the multi-response categories dichotomized. (Note: the set of categorical endpoints are: sex, race [dichotomized as white/nonwhite], ethnicity [dichotomized as 'Hispanic or Latino' or not].

# 3.9.2 Medical History

Medical history will be coded using MedDRA version 19.1 (or higher). The coded Preferred Terms (PT) will be summarized by treatment group and overall for the mITT Population. A subject will be counted only once for each preferred term. The summary will present the results alphabetically by System Organ Class (SOC) and, within SOC, by decreasing frequency for the Preferred Terms (PT).

# 3.93 Myasthenia Gravis History

The following gMG disease history data will be summarized by treatment group and overall for the mITT Population.

- Age at onset (years)
- Duration of disease (years)
  - = (Date of Study Day 1 Date of Diagnosis)/(365.25)


RA101495-02.201

Statistical Analysis Plan

Note: If the Date of Diagnosis day and month are missing impute July 2<sup>nd</sup>, if only the day is missing impute the 15<sup>th</sup>. If the imputed Date of Diagnosis date is later than the date of Study Day 1, impute Study Day 1.

- Symptoms at onset (Ocular/Generalized)
- MGFA Disease Class at Screening (Class II, III, or IV)
- Ever had a Crisis (Yes/No)
- Time since most recent crisis (months)

Mote: If the Date of Crisis day and month are missing impute July 2<sup>nd</sup>, if only the day is missing impute the 15<sup>th</sup>. If the imputed Date of Crisis date is later than the date of Study Day 1, impute the date of Study Day 1 st Recent Crisis Intervention Required (Hospitalized) uly members have MG (Yes, No) there of Family mem<sup>1</sup>

- Most Recent Crisis Intervention Required (Hospitalization, ICU, Tracheostomy)
- Family members have MG (Yes, No)
- Number of Family members with MG
- Closest relation with MG (Parent, Sibling, Child, Other) note: more than 1 relation may be selected
- Diagnosed with Thymoma (Yes, No)
- Prior Thymectomy (No: Yes [Total Thymectomy, Subtotal Thymectomy])
- Time from Thymectomy (months)
  - o Time since thymectomy will be calculated as (Date of Study Day 1 Date of Thymectomy)/(365.25/12)

Note: If the Date of Thymectomy day and month are missing impute July 2<sup>nd</sup>, if only the day is missing impute the 15<sup>th</sup>. If the imputed Date of Thymectomy date is later than the date of Study Day 1 impute the date of Study Day 1.

Additionally, a categorical summary of the age at disease onset overall and by gender will be performed by treatment group and overall.

### 3.10 Prior and Concomitant Medications

Prior and concomitant medications will be coded using WHO Drug (Version: v.2017JUN01 DDE B2 (enhanced)) and summarized by treatment group and overall for the Safety Population. MG specific medication will be summarized and listed separately (see Section 3.11 below) and not included in these summaries.

preterred (generic) drug name for the Safety Po presented only once for each therapeutic class and for each presented tables will be created for the following study periods:

A. Prior medications:

Prior medications are those that started Incidence of prior and concomitant medication will be presented by treatment group, therapeutic class, and preferred (generic) drug name for the Safety Population. A subject is counted only once for each therapeutic class and for each preferred drug

Prior medications are those that started and stopped before the Baseline visit

Concomitant medications in the Main Portion of the study are those concomitant medications taken during the Main Portion of the study (up to,


RA101495-02.201

Statistical Analysis Plan

but not including Day 84), including those started before and ongoing at first

C. Concomitant Medications in the Main and Extension Portions:

Portion of the study are those and ongoing into the Extension Portion.

The summaries will be performed for the 0.1 mg/kg and 0.3 mg/kg dose groups separately and combined, summarizing concomitant medications occurring in both the Main Portion and Extension Portion based following groups:

Output

Description

Descr

- 0.3 mg/kg Group: The subjects in the Main Portion 0.3 mg/kg group and the subjects in the Extension Portion in the placebo-0.3 mg/kg group.
- Combined 0.1 and 0.3 mg/kg Group. Combining the 0.1 mg/kg and 0.3 mg/kg groups.

Results will be presented in the following time-frames:

Within the First 12 Weeks:

This will include concomitant medications in in the Main Portion for subjects receiving active treatment in the Main Portion and in the first 12 weeks of the Extension Portion for subjects who received placebo in the Main Portion.

Within the First 24 Weeks: This will include concomitant medications in the Main Portion or the first 12 weeks of the Extension Study Period for subjects receiving active treatment in the Main Portion.

The following definitions will be used:

- Prior medications are those that started and stopped before the Baseline visit
- Concomitant medications are all medications taken during the study period, including those started before and are ongoing at first dose.
  - Concomitant medication in the Main Portion of the study are those concomitant medications taken during the Main Portion of the study (up to, but not including Day 84), including those started before and ongoing at first dose.

 o Concomitant medication in the Extension Portion of the study are those concomitant medications taken during the Extension Potion of the study

July missing, and it is unclear as to concomitant, it will be assumed that it is

3.11 MG Specific Prior and Concomitant Medications

MG specific medication will be presented separately from the other prior and concomitant medications (for both tables and listings). An MG specific medication defined by the "indication" value on the Prior and Concomitant Medication of the Prior therapy for MG".

The following tables summarizing "reated based on the Secondary of

- 1) MG specific prior medications: MG specific prior medications are those that started prior to the Baseline visit
- 2) MG specific medications taken at baseline. MG specific medications taken at baseline are those where the subject was on the medication at baseline (i.e., start date on or prior to Day 1 and stop date on or after Day 1 [or ongoing]).

Where an MG medication start date is partially or fully missing, and it is unclear as to whether the medication is prior or taken at baseline, it will be assumed that it is taken at baseline.

Note that a patient's MG medication may be in both of these categories.

In addition, a listing of MG specific medications which change from baseline through Day E84 will be produced.

Additionally, the number and percentage of patients who are taking one or more of the sets of MG specific medications presented in Table 12 (i.e., Groups A-E) will be summarized using the same 2 sets of tables:

- 1) MG specific prior medications
- 2) MG specific medications taken at baseline.

**Table 12: List of MG Medication Groups** 

| Group | <b>Concomitant Medication</b> | Preferred Term |
|-------|-------------------------------|----------------|
| A | prednisone for MG | PREDNISONE |


RA101495-02.201

Statistical Analysis Plan

| | other corticosteroids for MG | TBD* |
|---|------------------------------|-----------------------|
| D | Azathioprine | AZATHIOPRINE |
| В | Mycophenolate | MYCOPHENOLATE MOFETIL |
| С | IV Ig | IMMUNOGLOBULINS NOS |
| | SC Ig | IMMUNOGLOBULINS NOS |
| | Cyclosporine | CICLOSPORIN |
| | Cyclophosphamide | CYCLOPHOSPHAMIDE |
| | Methotrexate | METHOTREXATE |
| D | Tacrolimus | TACROLIMUS |
| | Rituximab | RITUXIMAB |
| | other third line | TBD* |
| | immunosuppressants | |
| E | plasma exchange | ALL OTHER NON- |
| | | THERAPEUTIC PRODUCTS |
| 1 | | |

<sup>\*</sup> *TBD*: to be determined; a list of corresponding medications and preferred terms will be provided by RA prior to database lock.

## 3.12 Exposure to Study Treatment

Study drug will be provided in prefilled syringes for self-injection using weight bracketed dosing (i.e., subjects will be provided prefilled syringes containing fixed amounts of RA101495 based on their weight, and each fixed amount will cover a range of subject weights).

Prefilled syringes will be dispensed to each subject at each study visit, beginning on Day 1 of the Treatment Period.

Subjects will be provided with training and detailed instructions on the administration of study drug using the prefilled syringes and the injection device.

The location and time of the study drug administrations will be presented in the listings for those visits where this information is collected for the Safety Population.

### 3.13 Safety Analysis

CO

Safety analysis results will be presented using the Safety Population by dose group and overall.

For safety analyses, summary results for the 0.1 mg/kg and 0.3 mg/kg dose groups will be presented individually and also combining the two dose groups.


RA101495-02.201

Statistical Analysis Plan

Listings for all safety data will be presented.

#### 3.13.1 Adverse Events

ions of variations thereof. All AEs will be coded using the Medical Dictionary of Regulatory Activities (MedDRA) Version 20.0 and will be classified by MedDRA system organ class (SOC) and preferred term (PT). Analyses of AEs will be performed using the Safety Population.

Treatment emergent AEs (TEAEs) are defined as follows:

- An AE that occurs after treatment start that was not present at the time of treatment start; or
- An AE that increases in severity after treatment start, if the event was present at the time of treatment start.

#### TEAE Analyses:

The following are the set of TEAE summaries to be provided:

- A. Overall summary of Treatment Emergent Adverse Events
- **B.** Incidence of Treatment Emergent Adverse Events by System Organ Class and Preferred Term
- C. Incidence of Treatment Emergent Adverse Events by System Organ Class. Preferred Term, and Maximum Severity
- **D.** Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug
- E. Incidence of Treatment Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term

For these summaries, the number and percentage of subjects who experienced at least one of the TEAE as well as the number and percentage of subjects who experienced each specific SOC and PT will be presented by treatment group. The corresponding number of TEAEs will also be presented for the Overall Summary of TEAEs table.

For the presentation of TEAE incidences, the SOCs will be sorted alphabetically, and within SOC, the preferred term (PT) will be used and presented by decreasing total frequency based on the total population.

For the overall summary of TEAEs, the following information will be provided

- Number of subjects with TEAEs
- Number of subjects with TEAE of Grade 2 or higher
- Number of subjects with a drug related TEAE
- Number of subjects with a TEAE leading to study discontinuation
- Number of subjects with an SAE.

For reporting, each TEAE will be assigned to either the Main Portion or the Extension Portion based on the AE start date:


RA101495-02.201

Statistical Analysis Plan

- If the start date of the TEAE is prior to Study Day 84 (i.e., the day the subject receives RA101495 in the Extension Portion) the TEAE will be assigned to
- The following are Study Period and Treatment Groups for which the set of TEAE analyses (listed as A-E above) will be performed.

  1. Main Portion:

  The set of TEAE analyses will be performed.

  The set of TEAE analyses will be performed.

### 2. Main Portion and Extension Portion:

This combines the Main Portion and the first 12 weeks of the Extension Portion. The set of TEAE analyses will be performed for the 0.1 mg/kg and 0.3 mg/kg dose groups separately and combined, summarizing TEAEs occurring in both the Main Portion and Extension Portion based on the following groups:

- 0.1 mg/kg Group: The subjects in the Main Portion 0.1 mg/kg group and the subjects in the Extension Portion in the placebo-0.1 mg/kg group.
- 0.3 mg/kg Group. The subjects in the Main Portion 0.3 mg/kg group and the subjects in the Extension Portion in the placebo-0.3 mg/kg group.
- Combined 0.1 and 0.3 mg/kg Group: Combining the 0.1 mg/kg and 0.3 mg/kg groups.

Results will be presented in the following time-frames:

- Within the First 12 Weeks: This will include AEs with a start date within the Main Portion for subjects receiving active treatment in the Main Portion and in the first 12 weeks of the Extension Portion for subjects who received placebo in the Main Portion.
- Within the 24 Weeks: This will include AEs with a start date in Main Portion or the first 12 weeks of the Extension Study Period for subjects receiving active treatment in the Main Portion.

Note: This is combining the RA101495 data from the Main Portion with the RA101495 data from the Extension Portion as described in Section 3.4.


#### 3.13.1.1 Treatment Emergent with Adverse Event Date Imputation

The following rules apply when determining if an AE is treatment-emergent in the If the year is the same as the year of the treatment start date, the day and month of the date of treatment start date will be assigned to the missing fields. If the year is prior to the year of the treatment start date, December 31 will be assigned to the missing fields. If the year is after the year of the date of the treatment start date, December 31 will be assigned to the missing fields. scenario where the start date is missing or partially missing. These rules provide an algorithm to "impute" a complete AE start date which will then be used to determine if the AE is treatment emergent.

## AE start date missing day and month:

- If the year is the same as the year of the treatment start date, the day and
- If the year is prior to the year of the treatment start date, December 31 will be
- If the year is after the year of the date of the treatment start date, January 1

#### AE start date missing month only:

The day will be treated as missing, and both month and day will be replaced according to the above procedure.

#### AE start date missing day only:

- If the month and year are the same as the month and year of the treatment start date, the day of the treatment start date will be assigned to the missing day.
- If either the year is before the year of the date of the treatment start date or if both years are the same, but the month is before the month of the treatment start date, the last day of the month will be assigned to the missing day.
- If either the year is after the year of the treatment start date or if both years are the same, but the month is after the month of the treatment start date, the first day of the month will be assigned to the missing day.

## AE start date completely missing:

- If the AE end date is complete and after the treatment start date, the treatment start date will be assigned to the missing start date.
- If the end date is complete and before the treatment start date, the end date will be assigned to the missing start date
- Otherwise the AE start date will be assigned the treatment start date.

The investigator should examination If the end date is complete and the imputed start date as above is after the end date, the start date will be imputed by the end date.

The investigator should assess the injection site (included as part of the physical examination) at each scheduled visit for:

- Pain, tenderness, erythema, and induration severity (Table 13)
  - o Erythema and induration: record the maximum linear diameter
- Blisters, ulceration, necrosis: record the maximum linear diameter and severity

 Lymphadenopathy

Table 13: Grading the Severity of Local Injection Site Reactions

| Local Reaction to<br>Injectable<br>Product | Grade 1<br>(Mild) | Grade 2<br>(Moderate) | Grade 3<br>(Severe) | Grade 4<br>(Potentially Life<br>Threatening) |
|---|---|---|---|---|
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever > 24 hours or<br>interferes with activity | Any use of narcotic<br>pain reliever or<br>prevents daily activity | Emergency room<br>visit or<br>hospitalization |
| Tenderness | Mild discomfort to touch | Discomfort with movement | Significant discomfort at rest | Emergency room<br>visit or<br>hospitalization |
| Erythema/<br>redness | 2.5 to 5.0 cm | 5.1 to 10.0 cm | > 10.0 cm | Necrosis or exfoliative dermatitis |
| Induration/<br>swelling | 2.5 to 5.0 cm and does not interfere with activity | 5.1 to 10.0 cm or interferes with activity | > 10.0 cm or prevents<br>daily activity | Necrosis |

Analysis of injection site reactions (ISRs) will include by treatment summaries of the following assessments using the subject's maximum grade over the corresponding study period as well as the number of times a grade was reported for a particular ISR.

• Any ISR, Pain, tenderness, erythema, and induration severity, and lymphadenopathy (categorical variables with grades 1 - 4, and absent).

This analysis will be performed for the:

- The Main Portion based on the Safety Population
- RA10495 Safety Population Within the First 12 Weeks: This will include RA10495 Safety Population Within the 24 Weeks: This will include ISRs with an assessment date in Main Portion or the first 12 weeks of the Extension Study Period for subjects receiving active treatment in the Main Portion.

  3.13.2 Clinical Laboratory Evaluation

  A list of the alignment of the a

Table 1.


RA101495-02.201

Statistical Analysis Plan

Quantitative laboratory endpoints will be summarized (including the value and change from baseline) at each scheduled assessment time point using descriptive statistics by dose group and combining the active dose groups for the Main Portion.

The liver functions test to be summarized via the National Cancer Institute (NCI)

Common Terminology Criteria for Adverse Events (CTCAE) criteria are provided in Table 14.

The number and percentage of subjects meeting these will be presented for the Main Portion to the O.1 and O.3 mg/kg does or the T

For the Extension Portion, active-dose results will be summarized for the scheduled visits based on the individual and combined 0.1 and 0.3 mg/kg dose groups as defined in Section 3.3 including results through 24 weeks of active-treatment.

Table 14: CTCAE Grading Criteria for Selected Liver Function Tests

| Lab Test | Grade/Criteria | | | |
|---|---|---|---|---|
| | 1 | 2 | 3 | 4 |
| alanine aminotransferase | > 1.0 - 3.0 | >3.0 5.0 | >5.0 - 20.0 | > 20.0 |
| (ALT) | (x ULN) | (x ULN) | (x ULN) | (x ULN) |
| alkaline phosphatase | >1.0 - 2.5 | >2.5 - 5.0 | >5.0 - 20.0 | > 20.0 |
| (ALP) | (x ULN) | (x ULN) | (x ULN) | (x ULN) |
| 11 | > 1.0 – 1.5 | >1.5 – 3.0 | >3.0 - 10.0 | > 10.0 |
| direct bilirubin | (x ULN) | (x ULN) | (x ULN) | (x ULN) |
| gamma-glutamyl | >1.0,2.5 | >2.5 - 5.0 | >5.0 - 20.0 | >20.0 |
| transferase | (x ULN) | (x ULN) | (x ULN) | (x ULN) |
| (GGT) | 00 | | | |
| Grading criteria based on Common Terminology Criteria for Adverse Events (CTCAE) v4.03 | | | | |

### 3.13.2.2 Pancreatic Enzymes: NCI CTCAE Grading

Amylase and lipase values will be summarized via the NCI CTCAE criteria provided in Table 15.

For the Extension Portion visits based on f The number and percentage of subjects meeting these criteria at each scheduled visit will be presented for the Main Portion by individual dose group and the combining

For the Extension Portion, active-dose results will be summarized for the scheduled visits based on for the combined 0.1 and 0.3 mg/kg dose groups as defined in Section 3.3 including results through 24 weeks of active-treatment.

Table 15: CTCAE Grading Criteria for Selected Pancreatic Enzyme Tests

| Lab Test | Grade/Criteria |
|--------------|----------------|
| CONFIDENTIAL | - |

#### RA101495-02.201

Statistical Analysis Plan

| | 1 | 2 | 3 | 4 | |
|---|---|---|---|---|---|
| 1 | > 1.0 – 1.5 | >1.5 – 2.0 | >2.0 - 5.0 | > 5.0 | |
| amylase | (x ULN) | (x ULN) | (x ULN) | (x ULN) | |
| limaga | > 1.0 – 1.5 | >1.5 – 2.0 | >2.0 - 5.0 | > 5.0 | Ç, |
| lipase | (x ULN) | (x ULN) | (x ULN) | (x ULN) | (O) |
| Grading criteria based on C | Common Terminology | Criteria for Adverse | Events (CTCAE) v4.0 | 03 | "VE, |
| 3.13.3 Vital Signs at Descriptive statistics pressure) values and assessment time point | for vital signs (in the change from | e., heart rate, bo | • • | and blood<br>ich scheduled | Walialions thereof. |
| 3.13.4 ECG | | | | " on Silv | |
| Descriptive statistics | for ECG parame | * | | nterval, QRS | |

### 3.13.3 Vital Signs and Other Physical Findings

#### 3.13.4 ECG

Descriptive statistics for ECG parameters (i.e., HR, PR interval, RR interval, QRS interval, QT interval, QTcB interval, and QTcF interval) at each assessment time point will be presented for the values and change from baseline scores by treatment group. QTc intervals will be calculated using both Fridericia's and Bazett's corrections.

Additionally, the ECG interpretation categorized as Normal, Abnormal – Clinically Significant, Abnormal – Not Clinically Significant, Not Evaluable, or Not Done will also be provided for each assessment time point (note: ECG interpretations of "Abnormal – Clinically Significant" would be recorded as AEs).

Note: ECG is not performed at Day 1, baseline values will be based on the Screening visit.

3.13.5 Physical Examination

The complete set physical examination findings will be provided in listings. Clinically significant physical examination abnormalities will be included and summarized as AEs if appropriate.

#### 3.14 Efficacy Analyses

Listings for all efficacy data will be presented.

# 3.14.1 Primary Efficacy Endpoint Analysis

For the primary efficacy endpoint, the change from baseline to Week 12 (Day 84) in Score Covariance a covariate.

The privo QM6 score, treatment group differences will be assessed by an Analysis of Covariance (ANCOVA) model, with treatment as a factor and baseline QMG score as

The primary efficacy analysis will be the comparison of the 0.3 mg/kg dose group versus the placebo dose group based on the ANCOVA model at a one-sided 0.10 significance level.

The comparison of the 0.1 mg/kg dose group versus the placebo dose group will be a secondary efficacy analysis tested at the 1-sided 0.10 level. Least-square means for


RA101495-02.201

Statistical Analysis Plan

each treatment group will also be presented. The following additional tests will be performed:

- A test for treatment effect pooling the 0.1 mg/kg and 0.3 mg/kg dose groups versus placebo: This will be performed by repeating the primary efficacy analysis ANCOVA with the 0.1 mg/kg, and 0.3 mg/kg dose groups with values of 0, mg/kg and 0.3 mg/kg dose groups versus placebo: This will be performed by repeating the primary efficacy analysis ANCOVA with the 0.1 mg/kg, and 0.3 mg/kg dose groups which is a superficient of the military of the mil • A test of linear trend across the 3 treatment groups: This will be performed by

The primary analysis population will be the mITT Population and LOCF is the primary method for handling missing data.

### 3.14.2 Secondary Efficacy Endpoints Analysis

The secondary efficacy endpoints are:

- Change from baseline to Week 12 in the MG-ADL scale
- Minimal symptom expression at Week 12, defined as an MG-ADL scale score of 0 or 1
- Change from baseline to Week 12 in the MG-Quality of Life 15r (MG-QOL15r)
- Change from baseline to Week 12 in the MG Composite
- A > 3-point reduction in OMG score at Week 12
- Requiring rescue therapy over the 12-week Treatment Period.

The secondary efficacy endpoints: Week 12 change from baseline in MG-ADL, MG-QOL15r, and MG Composite will be analyzed by an ANCOVA model similar to the primary efficacy endpoint analysis, with treatment as a factor and the corresponding baseline value as a covariate. Each of the active doses will be compared to the placebo group based on the ANCOVA model at the 1-sided 0.10 level.

For the categorical secondary endpoints: 'Minimal symptom expression at Week 12, defined as an MG-ADL scale score of 0 or 1', 'Subjects with > 3-point reduction in QMG score at Week 12' and 'Subjects requiring rescue therapy over the 12-week Treatment Period', the rate of subjects meeting the endpoint for each of the active treatment groups will be compared to the placebo group using a one-sided Fisher's exact test.

For the secondary endpoints the primary analysis population will be the mITT Population and LOCF is the primary method for handling missing data.


#### 3.15 Controlling for Multiplicity

This Phase 2 study will not control for multiple secondary endpoints.

### 3.15.1 Additional Analyses of Primary and Secondary Endpoints

The following are the set of additional analyses for the primary and secondary efficacy endpoint analyses:

- or variations thereof. a. The primary and secondary efficacy endpoint analyses will be performed on the PP population using the LOCF method.
- b. The primary and secondary efficacy endpoints will also be performed on the PP and mITT populations using the Observed Case analysis method (i.e., as defined in Section 3.2).
- c. The data from the placebo group Extension Portion (i.e., when the placebo group subjects are taking 0.1 mg/kg or 0.3 mg/kg RA101495) will be combined with the corresponding 0.1 mg/kg or 0.3 mg/kg RA101495 dose group data from the Main Portion following the method described in Section 3.4. Summary statistics will be provided for the values and change from baseline at each of the scheduled assessment time points for this combined data. These analyses will be done on the RA101495 Safety population. Note: no inferential analyses are planned. This analysis will be done for the change from baseline in QMG score and MG-ADL score using the LOCF methodology.
- d. The ANCOVA model as defined in Section 3.14.1 will be performed on the mITT Population using the LOCF method for missing data (as described in Section 3.2) including each of the following variables as an additional covariate (i.e., a separate ANCOVA model for each variable listed).
  - Sex (dichotomous class variable)
  - Age (continuous variable)
  - Duration of disease (continuous variable)
  - Age at disease onset (continuous variable)
  - Ever had a crisis(dichotomous yes/no class variable)
  - Prior thymectomy (dichotomous yes/no class variable)
  - Prior/current steroid therapy<sup>a</sup>
  - Prior/current immunosuppressive therapy (nonsteroidal)<sup>a</sup>
  - Prior history of intravenous or subcutaneous Immunoglobulin (IvIg) or (plasma exchange) PLEX
    - o Prior history of IvIg is defined in Concomitant Medications as "IMMUNOGLOBULINS NOS"; this is the ATC code via WhoDrug.
    - o Prior history of PLEX is defined in Concomitant Medications as "ALL OTHER NON-THERAPEUTIC PRODUCTS"; this is the ATC code via WhoDrug.

 a: Prior and concomitant medications will be reviewed and a list of those medications meeting this criteria will be finalized prior to database lock.

This analysis will be done for the change from baseline to Week 12 QMG score and MG-ADL score.

- e. For the Main Portion, the frequency distribution of the change from baseline will be summarized categorically for the following endpoints:
- Change from baseline to Week 12 in the MG-ADL scale levels from 0 to 15)

   Change from baseline to Week 12 in the MG-ADL scale (reduction baseline)

  - (reduction levels from 0 to 15)
  - Change from baseline to Week 12 in the MG Composite (reduction levels from 0 to 15)

Note: the tables may present reduction levels up to the maximum reduction level.

For each of these endpoints the number and % of subjects that have a reduction at a particular level and  $\geq$  that particular level (note: for these scales reduction from baseline indicates improvement) will be summarized. For each level a Fisher's exact test will be performed testing each active group versus the placebo group comparing the number of subjects with a change from baseline ≥ that particular level (and the combined active dose groups versus placebo).

These analyses will be done on the mITT population using the LOCF method.

Additionally, the data from the placebo group Extension Portion (i.e., when the placebo group subjects are taking 0.1 mg/kg or 0.3 mg/kg RA101495) will be combined with the corresponding 0.1 mg/kg or 0.3 mg/kg RA101495 dose group data from the Main Portion following the method described in Section 3.4. A summary of the change from baseline frequencies will be provided for the 0.1mg/kg and 0.3 mg/kg (and combined) dose groups.

These analyses will be done on the RA10495 Safety population using the LOCF method.

- A mixed model repeated measures (MMRM) analyzing the Main Portion. This analysis will be done on the following endpoints (i.e., a separate MMRM will be performed with each of these endpoints as the dependent variable):
  - Change from baseline in the QMG score
  - Change from baseline in the MG-ADL scale
  - Change from baseline in the MG-QOL15r survey

 • Change from baseline in the MG Composite

Based on the MMRM model, the treatment differences for each active dose group versus placebo as well as the treatment difference of the combined active doses versus placebo will be estimated for each of the post scheduled visits using LS means.

RM model will 1-

Mixed, example the support any manding at the support and support any manding at the support and support any manding at the support and support any manding at the support and su The MMRM model will be analyzed using SAS Proc Mixed, example SAS code for this MMRM is provided in the


RA101495-02.201

Statistical Analysis Plan

Appendix. This analysis will be performed on the mITT population using the LOCF Method and Observed Case Method for missing data (as described in Section 3.2).

- Atensions of variations thereof. g. An MMRM analyzing the data from both the Main Portion and first 12 weeks of the Extension Portion will be performed. This analysis will be done on the following endpoints (i.e., a separate MMRM will be performed with each of these endpoints as the dependent variable):
  - o Change from baseline in the QMG score
  - o Change from baseline in the MG-ADL scale
  - Change from baseline in the MG-OOL15r survey
  - Change from baseline in the MG Composite

Treatment, visit, treatment×visit interaction, and Study Portion, will be factors in the model and the corresponding baseline score will be a covariate (note: Study Portion is a categorical variable referring to the Main Portion and Extension Portion). For this analysis, the placebo subjects' Extension Study visit values will use the "matched" visits from the Main Portion. Specifically, the EXX visits (see Table 10) for the placebo subjects will map to Visit XX of the Main Portion (e.g., the Day E8 visit will map to Day 8 of the Main Portion). This has the Visits "matching" relative to the amount of time a subject has been on RA101495. For the extension period placebo data, the subject's baseline score (i.e., to be used when estimating change from baseline and used in the model as the baseline covariate) will be the Day 84 score.

The model will be adjusted for repeated measures using a within-subject unstructured covariance matrix (note: the covariance matrix structure may be simplified if there are convergence issues). The analysis will use the postbaseline scheduled visits (Day 8, 15, 29, 57, 84/E1, E8, E15, E29, E57, and E84).

Based on the MMRM model, the treatment difference of the combined active doses versus placebo will be estimated for each of the initial visits using LS means (Day 8, 15, 29, 57, and 84) and the LS-Means for the two active dose groups will be estimated for Visits: E1, E8, E15, E29, E57, and E84.

The MMRM model will be analyzed using SAS Proc Mixed, example SAS code for this MMRM is provided in the


RA101495-02.201

Statistical Analysis Plan

Appendix. This analysis will be performed on the mITT population using the LOCF Method and Observed Case Method for missing data (as described in Section 3.2).

extensions of variations thereof. h. The primary and secondary efficacy endpoint analyses will be performed on the mITT and PP population using the LOCF and Observed Case methods for the other scheduled assessment time points in the Main Portion.

#### 3.15.2 Pharmacodynamic Endpoints Analysis

Pharmacodynamic analyses will be performed on the PD Population.

The pharmacodynamic endpoints include:

- Sheep red blood cell (sRBC) lysis assay
- C5 levels

Summary statistics will be provided for the values, change from baseline, and percent change from baseline at each of the scheduled assessment time points.

For the Main Portion, the change from baseline for each of these endpoints will be assessed by an ANCOVA model with treatment as a factor and the corresponding baseline value as a covariate. Each of the active doses will be compared to the placebo group based on the ANCOVA model.

Additionally, the data from the placebo group Extension Portion (i.e., when the placebo group subjects are taking 0.1 mg/kg or 0.3 mg/kg RA101495) will be combined with the corresponding 0.1 mg/kg or 0.3 mg/kg RA101495 dose group data from the Main Portion following the method described in Section 3.4. Summary statistics will be provided for the values, change from baseline, and percent change from baseline at each of the scheduled assessment time points for this combined data.

These analyses will be performed on the PD population using observed cases (i.e., no censoring or imputation of data).

### 3.15.3 Pharmacokinetic Endpoints Analysis

Pharmacokinetic analyses will be performed on the PK Population.

The following pharmacokinetic endpoints will be presented in listings and summarized in tables.

- Plasma concentrations of RA101495 and its two major metabolites
- Maximum plasma concentration (C<sub>max</sub>)
- Time corresponding to  $C_{max}$  ( $t_{max}$ )
- Ratio of parent to metabolites (i.e., 2 metabolites).

These analyses will be performed on the PK population using observed cases (i.e., no censoring or imputation of data). Note: the PK parameters will be calculated by an external vendor and provided to PRA.


RA101495-02.201

Statistical Analysis Plan

#### 3.15.4 Exploratory Endpoints Analysis

For the functional sub-scores of the QMG, MG-ADL, QOL, and Composite scores Mechanistic biomarkers pertinent to MG pathophysiology [e.g., complement fixation, complement function, complement pathway proteins, autoantibody characterization (titer and immunoglobulin class) and inflammatory and confirmatory assay will be summarized for points. (defined in Section 3.7) the endpoints will be summarized using descriptive statistics at each scheduled assessment time point. Additionally, an ANCOVA model, with treatment as a factor and corresponding baseline score as a covariate will be performed to assess treatment group differences. This will be performed on the mITT population using LOCF.

The following exploratory endpoints will be summarized using descriptive statistics at each scheduled assessment time point in the Main Portion:

Pharmacogenomic analyses (optional) data collected will be presented in a listing.

### 3.16 Additional Analyses

### 3.16.1 Rescue Therapy

Subjects requiring rescue therapy over the 12-week Treatment Period is a secondary efficacy endpoint, with the analysis described in Section 3.14.2.

In addition to the secondary efficacy analyses the following analyses will be performed for the Main Portion on the mITT Population:

For those subjects who receive rescue therapy during the Main Portion, the time to rescue therapy will be summarized using descriptive statistics, including the number and percentage of subjects receiving rescue therapy, and time to rescue therapy. Time to rescue therapy (in days), will be calculated as:

Time to rescue therapy = (Date of Day 1 visit – Date of Rescue Therapy + 1)

The frequency and type of rescue medication (Immunoglobulin or Plasma Exchange) a subject receives will be summarized.

These summaries will be provided by dose group and for the 0.1 and 0.3 mg/kg dose groups combined.

For those subjects who receive rescue therapy while on RA101495 (i.e., both in the Main Portion and the first 12 weeks of the Extension Portion) the following summaries will be performed on the RA101495 Safety population:

The number and percentage of subjects receiving rescue therapy


RA101495-02.201

Statistical Analysis Plan

- The time from first dose of RA101495 to rescue therapy (summarized for those subjects who received rescue therapy)

No interim analysis is planned for the Main Portion of the study. Interim analyses of the Extension Portion of the study will be performed.

3.18 Timing of Primary Analysis

For the primary analyses of the Main Portion of the study will be performed. will be "frozen" and the set of primary, secondary, and a subset of the additional efficacy analysis will be performed in addition to a subset of the safety analyses corresponding to the Main Portion of the study.

3.19 Sample Size Considerations

For the primary efficacy endpoint, change from baseline to Week 12 (Day 84) in QMG score, assuming a difference in treatment group means of 4.5, an SD of 5.0, and 12 subjects per group, the study has approximately 81% power to detect a difference between an active and placebo treatment group based on a 1-sided t-test with a 0.10 type I error rate.

### 3.20 Replacement of Subjects

Subjects who prematurely discontinue participation prior to the Day 84 visit may be replaced in order to obtain at least 12 evaluable subjects per treatment arm.

### 3.21 Protocol Violations

a blinded 1 presented. Protocol violations will be assessed as major or minor prior to database unblinding, in a blinded manner. A listing of protocol violations by treatment group will be

## References

Barohn RJ, McIntire D, Herbelin L, Wolfe GI, Nations S, Bryan WW. Reliability testing of the quantitative myasthenia gravis score. Ann N Y Acad Sci. 1998;841:769-772.


RA101495-02.201

Statistical Analysis Plan

Benatar M, Sanders DB, Burns TM, Cutter GR, Guptill JT, Baggi F, et al; Task Force on MG Study Design of the Medical Scientific Advisory Board of the Myasthenia or variations thereof. Gravis Foundation of America. Recommendations for myasthenia gravis clinical trials. Muscle Nerve. 2012;45(6):909-917.

Burns, TM, Grouse CK, Conway MR, Sanders DB, and MG Composite and MG-QOL 15 study group. Construct and concurrent validation of the MG-QOL 15 in the practice setting. Muscle Nerve. 2010;41(2):219-226.

Burns TM, Sadjadi R, Utsugisawa K, Gwathmey KG, Joshi A, Jones S, et al.International clinimetric evaluation of the MG-QOL15, resulting in slight revision and subsequent validation of the MG-QOL15r. Muscle Nerve. 2016;54(6):1015-1022.

Katzberg HD, Barnett C, Merkies IS, Bril V. Minimal clinically important difference in myasthenia gravis: outcomes from a randomized trial. Muscle Nerve 2014;49(5):661-665.

Muppidi S, Wolfe GI, Conaway M, Burns TM; MG Composite and MG-QOL15 study group. MG ADL: still a relevant outcome measure. Muscle Nerve. 2011;44(5):727-731.

Sadjadi R, Conaway M, Cutter G, Sanders DB, Burns TM; MG Composite MG-QOL15 Study Group. Psychometric evaluation of the myasthenia gravis composite using Rasch analysis. Muscle Nerve. 2012;45(6):820-825.

profile

profile

profile

Inis document cannot be used to support any marker

This document cannot be used to support any marker Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. *Neurology*. 1999;52(7):1487-1489.

> 

## **Appendix 1: Sample SAS code for Repeated Measures Mixed Models**

The following is the sample code for the MMRM ANCOVA for the Main Portion described in Section 3.15.1, sub-section f. Note that this is an example to be used as a reference, the actual SAS code may differ from the sample provided below.

```
...e Study **;

...e Study **;

...e Study **;

...e Study **;

...e Study **;

...e study **;
  ** MMRM ANCOVA Code **;
  ** Analysis of Main Portion of the Study **;
 proc mixed data=XXXX;
** this data step subsets the LS means comparisons to within a visit, comparing against trt=0 **;

data diffs2;
   set diffs;
   where _trt=0 and visit=_visit;

run;

**

** MMRM ANCOVA Code

** Analysis of Main and Extense

** 1) for enhance.
 ** 1) for subjects randomized to treatment in main portion:
           visit x = visit
  ** 2) for subjects randomized to placebo in main portion:
            visit x = visit for main portion
  ** visit x = corresponding main portion visit for extension
 proc mixed data=simu4;
       class usubjid visit_x trt(Ref='0');
       model y_chg = y_base visit_x trt trt*visit_x/s;
       repeated /subject=usubjid type=UN;
       lsmeans visit x*trt/diff;
       ods output lsmeans=xlsmeans;
        ods output diffs=diffs;
              where visit in(8,15, 29, 57, 84, 91, 98, 112, 140, 167);
 run
          this data step subsets the LS means comparisons to within a
 visit, comparing against trt=0 **;
 data diffs2;
       set diffs;
      where trt=0 and visit x= visit x;
```


# **Appendix 2: Analyses Including Data After Day E84**

The following are the set of tables to summarize the data collected after Day E84. The tables will provide descriptive summary statistics (i.e., no inferential analyses will be performed).

#### 6.1 **Additional Analysis Population: Extension Population**

or variations thereof. The Extension Population will include all subjects who entered the Extension Period of the study as indicated by having a Day E1 visit.

### 6.2 Disposition

The Extension Period Disposition table will be amended to provide the number of subjects who completed Week E84 of the study and the reasons for discontinuation.

### Subject Switching From 0.1 mg/kg to 0.3 mg/kg

The date a subject in the 0.1 mg/kg group switched to 0.3 mg/kg (i.e., during the expansion phase of the study) will be presented in a listing.

Note: the date that a subject increased from the 0.1 mg/kg dose group to the 0.3 mg/kg dose group is recorded as "Date subject received first dose of open label study drug" in the eCRF form "Open Label Re-consent".

#### 6.4 Exposure

The number of years a patient is on the 0.1 mg/kg dose and 0.3 mg/kg dose group will be calculated for each subject using the following algorithm:

- The beginning of the interval will be the first day the subject begins that dose level. This will one of 3 timepoints:
  - o Day 1 of the Main Portion: the subject received this medication in the Main Portion)
    - Study Day 84/E1: the subject received placebo in the Main Portion and the dose of interest starting
  - The day the subject's dose increases from 0.1 mg/kg to 0.3 mg/kg: the subject was on 0.1 mg/kg and, during the Extension Period, the subject's dose was increased to 0.3 mg/kg.
- The end of the interval will be:
  - o The day the subject either discontinues or completes the study
  - o For the 0.1 mg/kg dose, the day prior to the subject taking the 0.3 mg/kg dose


RA101495-02.201

Statistical Analysis Plan

The number of years for a subject on zilucoplan will be calculated (for the 0.1 mg/kg and 0.3 mg/kg dose groups separately) as:

 $Interval = (date\ of\ end\ of\ Interval - date\ of\ beginning\ of\ interval)/365.25$ 

tensions of variations thereof. The total number of patient-years for a dose group will be the sum of the individual patient-years for that doses group within the corresponding population. This information will be presented in the adverse event table

### 6.5 Efficacy Endpoints

Efficacy endpoints will be summarized by the groups listed in Table 16.

**Table 16: Extension Table Groups** 

| Table Header | Treatment Group |
|-------------------|---------------------------------------------------------|
| Pbo/RA101495 | These are the subjects randomized Placebo in the Main |
| 0.1 mg/kg | Portion and randomized to 0.1 mg/kg in the Extension |
| | Portion |
| RA101495/RA101495 | These are the subjects randomized 0.1 mg/kg in the Main |
| 0.1 mg/kg | Portion and randomized to 0.1 mg/kg in the Extension |
| | Portion 4 dille |
| Pbo/RA101495 | These are the subjects randomized Placebo in the Main |
| 0.3 mg/kg | Portion and randomized to 0.3 mg/kg in the Extension |
| | Portion |
| RA101495/RA101495 | These are the subjects randomized 0.3 mg/kg in the Main |
| 0.3 mg/kg | Portion and randomized to 0.3 mg/kg in the Extension |
| | Portion |
| Total | These are all subjects in the population. |

Additional information for the efficacy tables:

- The analysis population for the tables will be the Extension Population (defined in Section 6.1)
- The endpoints will be summarized starting at Week E1 through Week E84 (i.e., the last scheduled visit for the study)
- The Observed Case method for the Extension Period, as described in Section 3.2.2, will be applied.
- The value and change from baseline values will be summarized. Baseline will

The efficacy endpoints to be summarized include the primary and secondary change from baseline efficacy endpoints (i.e., QMG, MG-ADL, MG-QOL15r, and MG Composite).


#### 6.6 Safety Endpoints

#### 6.6.1 Adverse Events

extensions of variations thereof. TEAEs will be summarized across the entire study, excluding TEAEs occurring during the Main Portion of the study for those subjects on placebo during the Main Portion. Results will be summarized by the dose the subject was on (i.e., 0.1 mg/kg or 0.3 mg/kg) at the start date of the TEAE as well as "Overall".

The AE tables will include:

- TEAEs by SOC/PT
- Related TEAEs by SOC/PT
- Serious TEAEs by SOC/PT

In addition, an overall summary of TEAEs table will present the following:

- Any TEAEs
- Any Grade 2 or Greater, Grade 3 or Greater, and Grade 4 or Greater, TEAEs
- Any Treatment-Related TEAEs
- Any Grade 2 or Greater, Grade 3 or Greater, and Grade 4 or Greater, Treatment-Related TEAEs
- Any TEAEs with Outcome of Death
- Any Serious TEAEs
- Any Treatment-Related Serious TEAE

The AE, SAE, and TEAEs with an outcome of Death listings will be updated to include the dose the subject is on at the start of the event. As the subject-years exposure will be notably different between the 0.1 mg/kg group and the 0.3 mg/kg group a footnote will be provided to provide context to the AE frequencies and percentages. The subject-years will be calculated using the method described in Section 6.3.

For each of these AE tables the total number of patient-years for each treatment group (and overall) as defined in Section 6.3 will be presented.

#### Labs and Vital Signs 6.6.2

Labs and vital sign endpoints will be summarized in the same manner as the efficacy endpoints (defined in Section 6.5).

